# Johnson & Johnson Vision Care, Inc.

# Clinical Study Protocol

Title: Design Validation of senofilcon A with New UV-blocking Additive

Protocol: CR-6305

Version: 4.0, Amendment 3.0

Date: 14 November 2018

Investigational Products: ACUVUE OASYS $^{\otimes}$  with Transitions $^{TM}$  Light Intelligent Technology $^{TM}$ 

Key Words: senofilcon A, ACUVUE OASYS®, ACUVUE OASYS with Transitions Light Intelligent Technology, daily wear reusable, dispensing

# Statement of Compliance to protocol, GCP and applicable regulatory guidelines:

This trial will be conducted in compliance with the protocol, ISO 14155, the International Conference on Harmonization Good Clinical Practice E6 (ICH-GCP), the Declaration of Helsinki, and all applicable regulatory requirements.

## **Confidentiality Statement:**

This document contains confidential information, which should not be copied, referred to, released or published without written approval from Johnson & Johnson Vision Care, Inc. The information may not be disclosed to others except to the extent necessary to obtain Institutional Review Board/Independent Ethics Committee approval and informed consent, or as required by International, Federal and State Laws, as applicable. Persons to whom this information is disclosed must be informed that this information is privileged and confidential and that it should not be further disclosed without the written permission of Johnson & Johnson Vision Care, Inc. Any supplemental information that may be added to this document is also confidential and proprietary to Johnson & Johnson Vision Care, Inc. and must be kept in confidence in the same manner as the contents of this document.

# TABLE OF CONTENTS

| DDOTOCOL TITLE MIL | MDED VEDSION | 6 |
|---|---|---|
| | MBER, VERSION | |
| | ADDRESS | |
| | TURES | |
| | AND BACKGROUND | |
| | riptions of Investigational Products | |
| | Investigational Products | |
| | dings from Nonclinical Studies | |
| | own Risks and Benefits to Human Subjects | |
| | ure References and Prior Clinical Data Relevant to Pr | |
| • | TEG ENDRODITE AND INDOTHEGES | |
| | 'ES, ENDPOINTS AND HYPOTHESES | |
| 1 | ~ ¬ 1 · | |
| | ficacy Endpoints: | |
| | fety Endpoints: | |
| • | Endpoints: | |
| • | oints: | |
| • 1 | | |
| | potheses | |
| • | Hypotheses | |
| 3. TARGETED STUD | Y POPULATION | 20 |
| 3.1. General Charact | teristics | 20 |
| 3.2. Inclusion Criteri | ia | 21 |
| 3.3. Exclusion Criter | ria | 21 |
| 3.3.1. Systemic M | ledications | 22 |
| 3.4. Enrollment Strat | tegy | 23 |
| 4. STUDY DESIGN A | ND RATIONALE | 23 |
| 4.1. Description of S | tudy Design | 23 |
| 4.2. Study Design Ra | ationale | 24 |
| 4.3 Enrollment Targ | get and Study Duration | 24 |

| 5. TE | EST ARTICLE ALLOCATION AND MASKING | 24 |
|-------|-----------------------------------------------------|----|
| 5.1. | Test Article Allocation | 24 |
| 5.2. | Masking | 25 |
| 5.3. | Procedures for Maintaining and Breaking the Masking | 25 |
| 6. ST | TUDY INTERVENTION | 26 |
| 6.1. | Identity of Test Articles | 26 |
| 6.2. | Ancillary Supplies/Products | 26 |
| 6.3. | Administration of Test Articles | 26 |
| 6.4. | Packaging and Labeling | 27 |
| 6.5. | Storage Conditions | 27 |
| 6.6. | Collection and Storage of Samples | 27 |
| 6.7. | Accountability of Test Articles | 27 |
| 7. ST | TUDY EVALUATIONS | 28 |
| 7.1. | Time and Event Schedule | 28 |
| 7.2. | Detailed Study Procedures | 29 |
| V | SIT 1 | 29 |
| V | SIT 2 | 34 |
| FI | NAL EVALUATION | 35 |
| 7.3. | Unscheduled Visits | 36 |
| 7.4. | Laboratory Procedures | 37 |
| 8. SU | JBJECTS COMPLETION/WITHDRAWAL | 37 |
| 8.1. | Completion Criteria | 37 |
| 8.2. | Withdrawal/Discontinuation from the Study | 37 |
| 9. PF | RE-STUDY AND CONCOMITANT INTERVENTION/MEDICATION | 38 |
| 10. | DEVIATIONS FROM THE PROTOCOL | 38 |
| 11. | STUDY TERMINATION | 38 |
| 12. | PROCEDURE FOR HANDLING PRODUCT QUALITY COMPLAINTS | 39 |
| 13. | ADVERSE EVENTS | 40 |
| 13.1. | Definitions and Classifications | 40 |
| 13.2. | Assessing Adverse Events | 42 |
| 13 | .2.1. Causality Assessment | 43 |
| | .2.2. Severity Assessment | |
| 13.3. | Documentation and Follow-Up of Adverse Events | 43 |
| 13 / | Reporting Adverse Events | 15 |

| 13 | .4.1. Reporting Adverse Events to Sponsor | 45 |
|---|---|---|
| 13 | .4.2. Reporting Adverse Events to the Responsible IEC/IRB and Health Authorit | ies46 |
| 13 | .4.3. Event of Special Interest | 46 |
| 13.5. | Reporting of Pregnancy | 46 |
| 14. | STATISTICAL METHODS | 46 |
| 14.1. | General Considerations | 46 |
| 14.2. | Sample Size Justification | 47 |
| 14.3. | Analysis Populations | 51 |
| 14.4. | Level of Statistical Significance | 51 |
| 14.5. | Primary Analysis | 51 |
| 14.6. | Secondary Analysis | 56 |
| 14.7. | Other Exploratory Analyses | 56 |
| 14.8. | Interim Analysis | 56 |
| 14.9. | Procedure for Handling Missing Data and Drop-Outs | 57 |
| 14.10 | ). Procedure for Reporting Deviations from Statistical Plan | 57 |
| 15. I | DATA HANDLING AND RECORD KEEPING/ARCHIVING | 57 |
| 15.1. | Electronic Case Report Form/Data Collection | 57 |
| 15.2. | Subject Record | 57 |
| 16. I | DATA MANAGEMENT | 58 |
| 16.1. | Access to Source Data/Document | 58 |
| 16.2. | Confidentiality of Information | 58 |
| 16.3. | Data Quality Assurance | 58 |
| 17. I | MONITORING | 59 |
| 18. I | ETHICAL AND REGULATORY ASPECTS | 59 |
| 18.1. | Study-Specific Design Considerations | 59 |
| 18.2. | Investigator Responsibility | 59 |
| 18.3. | Independent Ethics Committee or Institutional Review Board (IEC/IRB) | 60 |
| 18.4. | Informed Consent | 61 |
| 18.5. | Privacy of Personal Data | 61 |
| 19. | STUDY RECORD RETENTION | 62 |
| 20. I | FINANCIAL CONSIDERATIONS | 63 |
| 21. I | PUBLICATION | 63 |
| 22. I | REFERENCES | 63 |
| APPEN | IDIX A: PATIENT REPORTED OUTCOMES (STUDY QUESTIONNAIRES) | 65 |

| APPENDIX B: PATIENT INSTRUCTION GUIDE | 72 |
|---|---|
| APPENDIX C: PACKAGE INSERT (APPROVED PRODUCT) | 73 |
| APPENDIX D: | 76 |
| LENS FITTING CHARACTERISTICS | |
| SUBJECT REPORTED OCULAR SYMPTOMS/PROBLEMS | 84 |
| , FRONT AND BACK SURFACE LENS DEPOSIT GRADING PROCED | URE 86 |
| DETERMINATION OF DISTANCE SPHEROCYLINDRICAL REF | RACTIONS |
| BIOMICROSCOPY SCALE | 99 |
| KERATOMETRY PROCEDURE | 105 |
| DISTANCE AND NEAR VISUAL ACUITY EVALUATION | 107 |
| DISTANCE LOGMAR VISUAL ACUITY MEASUREMENT PROCED | URE112 |
| , PATIENT REPORTED OUTCOMES | |
| , WHITE LIGHT LENS SURFACE WETTABILITY | 118 |
| VISUAL ACUITY CHART LUMINANCE AND ROOM ILLUMINESTING. | MINATION |
| PROTOCOL COMPLIANCE INVESTIGATOR(S) SIGNATURE PAGE | 128 |
| TABLE OF CONTENTS Figure 1: Study Flowchart | 13 |
| TABLE OF CONTENTS | |
| Table 1: Disallowed systemic medications (less than one year of continual use) | |
| Table 2: Test Articles | |
| Table 3: Ancillary Supplies | |
| Table 5: Historical Studies Included in Sample Size Calculation | |
| Table 8: Descriptive Summary of Mechanical Lens Fitting Pooled Across all Histor | |
| Table 9: Descriptive Summary of Slit Lamp Findings Pooled Across all Historical Stu | 48<br>idies 48 |
| Table 11: Sample Size Estimates and Power Calculations for Primary Endpoints Table 12: Sample Size Estimates and Power Calculations for Secondary Endpoints | |

# PROTOCOL TITLE, NUMBER, VERSION

Title: Design Validation of senofilcon A with New UV-blocking Additive

Protocol Number: CR-6305 Version: 4.0, Amendment 3.0 Date: 14 November 2018

#### SPONSOR NAME AND ADDRESS

Johnson & Johnson Vision Care, Inc. (JJVCI) 7500 Centurion Parkway Jacksonville, FL 32256

## **MEDICAL MONITOR**

Name: John R. Buch, O.D., M.S., F.A.A.O. Title: Senior Principal Research Optometrist

Address: 7500 Centurion Parkway, Suite 100, Jacksonville, FL 32256

Email: jbuch@its.jnj.com

The Medical Monitor must be notified by the clinical institution/site by e-mail, fax, or telephone within 24 hours of learning of a Serious Adverse Event. The Medical Monitor may be contacted during business hours for adverse event questions. General study related questions should be directed towards your assigned clinical research associate.

The Medical Monitoring Plan is maintained as a separate document and included in the Trial Master File.

## **AUTHORIZED SIGNATURES**

The signature below constitutes the approval of this protocol and the attachments, and provides the necessary assurances that this trial will be conducted according to all stipulations of the protocol, including all statements regarding confidentiality, and according to local legal and regulatory requirements and applicable U.S. federal regulations,<sup>4</sup> ICH guidelines,<sup>2</sup> ISO 14155,<sup>1</sup> and the Declaration of Helsinki.<sup>3</sup>

| Author / Study | Can Electronia Signatura Domant | |
|---|---|---|
| Responsible Clinician | See Electronic Signature Report John R. Buch, O.D., M.S. | DATE |
| | Senior Principal Research Optometrist, JJVCI | DITTE |
| Clinical Operations | | |
| Manager | See Electronic Signature Report | DATE |
| | Clinical Operations Manager, JJVCI | DATE |
| Biostatistician | See Electronic Signature Report | DATE. |
| | Biostatistician II, JJVCI | DATE |
| Biostatistician | See Electronic Signature Report | |
| Reviewer | Sr. Manager, Biostatistics JJVCI | DATE |
| Data Management | See Electronic Signature Report | DATE |
| | Clinical Project Manager – Data & Systems,<br>JJVCI | DATE |
| Reviewer | See Electronic Signature Report | |
| | Clinical Research Fellow, JJVCI | DATE |
| Approver | See Electronic Signature Report | |
| | Dir. Sphere - Light Management - Lens care, JJVCI | DATE |

# **CHANGE HISTORY**

| Version | Originator | Description of Change(s) and Section<br>Number(s) Affected | Date |
|---|---|---|---|
| 1.0 | John R. Buch | Original Protocol | 06 September 2018 |
| 2.0 | John R. Buch | Amendments to make more compliant to ISO11980: 1. Added exclusion criteria of herpetic keratitis and pathological dry eye 2. Baseline ocular physiological findings must be Grade 0 or 1. Amendment recommended by IRB: 1. Include vitamin A analogs to Table 1. Clarified logMAR acuity room illumination, chart luminance, and which eye will read which chart. | 19 September 2018 |
| 2.0 | I-1 - D D - 1 | | 00.0-4-12010 |
| 3.0 | John R. Buch | <ul> <li>Amendments to V2 include: <ul> <li>Clarified temporary use of suspect medications in Section 3.3.1.</li> <li>Section 7.2: Visit 2 occurs 13-15 days following Visit 1.</li> <li>Section 7.2: added applicable for logMAR visual acuity</li> </ul> </li> <li>Updated medication spelling errors</li> <li>Table 1: Inserted study specific labels</li> </ul> | 08 October 2018 |
| 4.0 | | <ol> <li>Updated verbiage in Hypotheses <ul> <li>3 and 4 to match the acceptance criteria in the Customer</li> <li>Requirement Document (VIS-Dval-000194/4) dated on August 29, 2018.</li> </ul> </li> <li>Added details to the sample size justification in section 14.3.</li> <li>Updated the hypotheses 3 and 4 (null and alternative) in Section 14.</li> </ol> | 14 November 2018 |

# **SYNOPSIS**

| Protocol Title | Design Validation of senofilcon A with New UV-blocker<br>Additive |
|---|---|
| Sponsor | JJVCI, 7500 Centurion Parkway, Jacksonville, FL 32256 |
| Clinical Phase | Design input validation |
| Trial Registration | This study will be registered on ClinicalTrials.gov by the Sponsor |
| Test Article(s) | Investigational Products: senofilcon A with new UV-blocking additive (i.e., ACUVUE OASYS with Transitions Light Intelligent Technology). Control Products: senofilcon A without new UV-blocking additive (i.e., ACUVUE OASYS®). |
| Wear and Replacement | Wear Schedule: daily wear |
| Schedules | Replacement Schedule: 2 weeks |
| Objectives | The primary purpose of this randomized study is to demonstrate that the 4GT Test lens senofilcon A with new UV-blocker, in its final lens design ECL600, meets the design validation requirements related to overall CLUE comfort, logMAR visual acuity, quality of vision in bright light, eye health, and fit acceptance. |
| Study Endpoints | Primary endpoints: logMAR visual performance, slit lamp findings (Graded 3 or higher), fit acceptance, overall CLUE comfort and satisfaction of vision in bright light. |
| | Secondary endpoints: CLUE handling and CLUE overall quality of vision. |
| Study Design | This is a 2-visit, multi-site, partially subject-masked, 2-arm parallel, controlled, randomized and dispensing trial. Subjects will be randomized to one of two study lenses for the entire duration of the study. The study lenses will be worn for a period of 2 weeks each in a bilateral fashion. Subjects will be advised to wear the study lens for a minimum of 5 days per week for at least 6 hours per day. See the flow chart at the end of the synopsis table for the schematic of the study visits and procedures of main observations (Figure 1Figure 1). |
| Sample Size | Multiple external investigational sites will enroll approximately |
| Sample Size | 236 subjects with the intent of completing approximately 224. |
| Study Duration | The study is approximately two weeks per subject. The enrollment period is approximately two weeks, resulting in a |

| | total study duration of approximately four weeks from first subject first visit to last subject last visit. |
|---|---|
| Anticipated Study<br>Population | Healthy adult males and females of any race and ethnicity will<br>be recruited. All subjects will be habitual wearers of spherical<br>soft contact lenses. |
| Eligibility Criteria (Inclusion) | <ol> <li>Potential subjects must satisfy all of the following criteria to be enrolled in the study: <ol> <li>The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.</li> <li>Appear able and willing to adhere to the instructions set forth in this clinical protocol.</li> <li>Between 18 and 49 (inclusive) years of age at the time of informed consent.</li> <li>Eligible presbyopes will be those that wear full distance contact lenses in both eyes, then wear reading glasses over them when needed for near vision.</li> </ol> </li> <li>The subject is a current spherical soft contact lens wearer in both eyes with a minimum of 6 hours/day and 5 days/week wear time over the last 30 days by self-report.</li> <li>Subjects must be able and willing to wear the study lenses at least 6 hours a day, a minimum of 5 days per week</li> <li>Subjects must own a wearable pair of distance spectacles.</li> <li>The subject's vertex-corrected spherical equivalent distance refraction must be in the range of -1.00 to -6.00 D (inclusive) in each eye.</li> <li>The subject's refractive cylinder must be 0.00 to -1.00 D (inclusive) in each eye.</li> <li>The subject must have a spherocylindrical best corrected distance Snellen visual acuity of 20/25<sup>+3</sup> or better in each eye.</li> </ol> |
| Eligibility Criteria (Exclusion) | <ol> <li>Potential subjects who meet any of the following criteria will be excluded from participating in the study:</li> <li>Currently pregnant or lactating (subjects who become pregnant during the study will be discontinued).</li> <li>Any active or ongoing systemic disease (e.g., Sjögren's Syndrome), infectious disease (e.g., hepatitis, tuberculosis), contagious immunosuppressive diseases (e.g., HIV), autoimmune disease (e.g. rheumatoid arthritis).</li> <li>Subjects taking suspect oral medications for less than one year. (See Section 3.3.1 for suspect medications and more details).</li> <li>Any prescribed or over the counter (OTC) ocular medication.</li> </ol> |

| | <ol> <li>Any known hypersensitivity or allergic reaction to Optifree® PureMoist® multi-purpose care solution or Eye-Cept® rewetting drop solution.</li> <li>Toric, extended wear, monovision or multi-focal contact lens correction.</li> <li>Any previous or planned (during the course of the study) ocular surgery (e.g., PRK, LASIK, etc.).</li> <li>Participation in any contact lens or lens care product clinical trial within 30 days prior to study enrollment.</li> <li>Participation in clinical trials involving the Test lens within 3 months prior to study enrollment.</li> <li>Employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician).</li> <li>Binocular vision abnormality or strabismus by self-report or prior medical history.</li> <li>History of recurrent corneal erosions, herpetic keratitis, or pathological dry eye.</li> <li>Any active ocular allergies, infections or other ocular abnormalities (entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma) that the investigator determines may interfere with the outcomes of this study or otherwise contraindicate participation in the study.</li> <li>Any Grade 2 or greater slit lamp findings (e.g., edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) on the FDA Slit Lamp Classification Scale.</li> <li>Any previous history or signs of a contact lens-related corneal inflammatory event (e.g., past peripheral ulcer or round peripheral scar) within the past 3 years of otherwise successful contact lens wear.</li> </ol> |
|---|---|
| Disallowed Medications/Interventions | Suspect oral medications listed in Section 3.3.1 taken for less than one year on a continual (year-round, routine) basis. Any prescribed or over the counter (OTC) ocular medication. |
| Measurements and Procedures | Monocular distance visual acuity on logMAR scale using ETDRS charts, physiological responses, fitting characteristics, individual performance item (CLUE subjective question), CLUE overall comfort, vision and handling. |
| Microbiology or Other<br>Laboratory Testing | The optical bench will be used to measure the light transmission characteristics for all worn Test lenses. The findings are for internal information only and will not be part of the final report. |
| Study Termination | The occurrence of one or more Unanticipated Adverse Device Effect (UADE), or any SAE where relationship to study agent cannot be ruled out, will result in stopping further dispensing investigational product. In the event of a UADE or SAE, the Sponsor Medical Monitor may unmask the treatment regimen |

| | of subject(s) and may discuss this with the Principal Investigator before any further subjects are enrolled. |
|---|---|
| Ancillary Supplies/ Study-<br>Specific Materials | Opti-Free® PureMoist® and preservative free rewetting drops/artificial tears |
| Principal Investigator(s) and Study Institution(s)/Site(s) | A full list of Principal Investigators, clinical sites, and institutions is kept separately from the Study Protocol and is included in the study Trial Master File. |

Figure 1: Study Flowchart



# COMMONLY USED ABBREVIATIONS AND DEFINITIONS OF TERMS

ADD Plus Power Required for Near Use

ADE Adverse Device Effect

AE Adverse Event/Adverse Experience
BCVA Best Corrected Visual Acuity

BSCVA Best Spectacle Corrected Visual Acuity

CFR Code of Federal Regulations
CLUE Contact Lens User Experience

COAS Complete Ophthalmic Analysis System

COM Clinical Operations Manager
CRA Clinical Research Associate
CRD Customer Requirement Document

CRF Case Report Form

CRO Contract Research Organization

CT Center Thickness

CTP Clinical Technical Procedure

D Diopter

DMC Data Monitoring Committee eCRF Electronic Case Report Form EDC Electronic Data Capture

ETDRS Early Treatment Diabetic Retinopathy Study

FDA Food and Drug Administration

GCP Good Clinical Practice

HIPAA Health Insurance Portability and Accountability Act

IB Investigator's Brochure ICF Informed Consent Form

ICH International Conference on Harmonization

IDEInvestigational Device ExemptionIECIndependent Ethics CommitteeIPPIndividual Patient ProfilesIRBInstitutional Review Board

ISO International Organization for Standardization

ITT Intent-to-Treat

JJVCI Johnson & Johnson Vision Care, Inc.

LC Limbus Center

LogMAR Logarithm of Minimal Angle of Resolution MedDRA<sup>©</sup> Medical Dictionary for Regulatory Activities

MOP Manual of Procedures

NIH National Institutes of Health

OD Right Eye

OHRP Office for Human Research Protections
OHSR Office for Human Subjects Research

OS Left Eve

OTC Over the Counter

OU Both Eyes

PD Protocol Deviation

PHI Protected Health Information

PI Principal Investigator
PIG Patient Instruction Guide
PQC Product Quality Complaint
PRO Patient Reported Outcome

QA Quality Assurance OC Quality Control

SAE Serious Adverse Event/Serious Adverse Experience

SAP Statistical Analysis Plan SAS Statistical Analysis System

SD Standard Deviation

SOP Standard Operating Procedure

UADE Unanticipated Adverse Device Effect

USADE Unanticipated Serious Adverse Device Effect

UV Ultraviolet VA Visual Acuity

## 1. INTRODUCTION AND BACKGROUND

Medical devices include everything from simple tongue depressors to contact lenses to complex programmable pacemakers. Global regulations and standards require medical device manufacturers to have a quality system for the design, manufacture, packaging, labeling, and storage of finished medical devices. As a result, JJVCI must have a quality system that complies with several sets of regulations and standards from around the globe:

- US: FDA Quality System Regulation 21 CFR Part 820
- Europe: MDD 93/42/EEC ISO 13485:2003 Quality management systems
- Japan: Japan MHLW Ministerial Ordinance 169, 2004
- Canada: Canadian Medical Device Regulations

The investigational product used in this study was FDA-approved in April 2018. The intent of this study is to validate that the product meets all quality system/design control requirements in accordance with federal regulations.

The Test and Control contact lenses used in this study are both manufactured with senofilcon A material – the Test lens will contain the new UV-blocker. The new UV-blocker darkens in the presence of ultraviolet (UV) and high energy visible (HEV) light and lightens in its absence. That is, it has photochromic properties. Since no other photochromic contact lens is commercially available, the choice of predicate device was based on the similarity of base material.

In addition to correcting myopia and hyperopia, the Test lens will attenuate bright light. The lens has been evaluated on over 1,000 subjects with an excellent safety profile as described in the Investigator's Brochure (IB).<sup>5</sup> It is intended for daily wear only and replaced every two weeks.

# 1.1. Name and Descriptions of Investigational Products

Test lens: ACUVUE OASYS with Transitions Light Intelligent Technology. This product is made with a version of senofilcon A that has been modified with the addition of the new UV-blocker.

Control lens: ACUVUE OASYS®. This product is also made with senofilcon A making the comparison to the Test lens as valid as possible.

The Test and Control lenses are otherwise made with the same with respect to overall lens diameter (14.0 mm) and base curve radius (8.4 mm). The Test lens is approximately 15 microns thicker in the center than the Control lens (0.85 vs. 0.70 mm, respectively). Further details about the test articles are found in Section 6 of this protocol.

# 1.2. Intended Use of Investigational Products

The intended use of the investigative product is for correcting myopia and for the attenuation of bright light. During the study, each study article will be worn bilaterally in daily wear, reusable modality for at least 6 hours per day, and at least 5 days per week. The subject will wear only one of the study lenses for two weeks.

# 1.3. Summary of Findings from Nonclinical Studies

All previous pre-clinical findings were deemed satisfactory prior to proceeding with clinical trials on humans. For the most comprehensive nonclinical information regarding ACUVUE OASYS Transitions refer to the latest version of the Investigator's Brochure.

#### 1.4. Summary of Known Risks and Benefits to Human Subjects

The benefits to the subject are the same for any contact lens, namely the correction of their refractive error, with the added benefit of the attenuation of bright light for those subjects randomized to wear the Test lens.

The risks to the subject are the same for any contact lens, namely those stated in the Informed Consent Form (ICF), with the added precaution that the Test lens should be worn on both eyes. Wearing only one photochromic lens may cause disturbances in motion perception when the lens is activated.

For the most comprehensive risk and benefit information regarding ACUVUE OASYS Transitions refer to the latest version of the Investigator's Brochure.

# 1.5. Relevant Literature References and Prior Clinical Data Relevant to Proposed Clinical Study

Prior clinical data is summarized in the Investigator's Brochure.

The literature is absent of any articles pertaining to soft contact lenses containing the new type of UV-blocker. A list of relevant literature references pertaining to glare, eyestrain, and light filtering is provided:

- 1. Agarwal, S., Goel, D., & Sharma, A. (2013). Evaluation of the factors which contribute to the ocular complaints in computer users. J Clin Diagn Res,7(2), 331-335.
- 2. Eperjesi, F., Fowler, C. W., & Evans, B. J. (2002). Do tinted lenses or filters improve visual performance in low vision? A review of the literature. Ophthalmic and Physiological Optics, 22(1), 68-77.
- 3. Hickcox, K. S., Narendran, N., Bullough, J. D., & Freyssinier, J. P. (2013). Effect of different coloured luminous surrounds on LED discomfort glare perception. Lighting Research and Technology, 1477153512474450.
- 4. Leguire, L. E., & Suh, S. (1993). Effect of light filters on contrast sensitivity function in normal and retinal degeneration subjects. Ophthalmic and Physiological Optics, 13(2), 124-128.
- 5. Morse, R. S. (1985, October). Glare filter preference: influence of subjective and objective indices of glare, sharpness, brightness, contrast and color. In Proceedings of the Human Factors and Ergonomics Society Annual Meeting(Vol. 29, No. 8, pp. 782-786). SAGE Publications.
- 6. Pérez-Carrasco, M. J., Puell, M. C., Sánchez-Ramos, C., López-Castro, A., & Langa, A. (2005). Effect of a yellow filter on contrast sensitivity and disability glare after laser in situ keratomileusis under mesopic and photopic conditions. Journal of Refractive Surgery, 21(2), 158-165.
- 7. Sheedy, J. E., Hayes, J., & ENGLE, J. (2003). Is all asthenopia the same? Optometry & Vision Science, 80(11), 732-739.
- 8. Steen, R., Whitaker, D., Elliott, D. B., & Wild, J. M. (1994). Age-related effects of glare on luminance and color contrast sensitivity. Optometry & Vision Science, 71(12), 792-796.
- 9. Vincent, A. J., Spierings, E. L., & Messinger, H. B. (1989). A controlled study of visual symptoms and eye strain factors in chronic headache. Headache: The Journal of Head and Face Pain, 29(8), 523-527.
- 10. Wilkins, A. J., & Evans, B. J. (2010). Visual stress, its treatment with spectral filters, and its relationship to visually induced motion sickness. Applied Ergonomics, 41(4), 509-515.

# 2. STUDY OBJECTIVES, ENDPOINTS AND HYPOTHESES

# 2.1. Objectives

## **Primary Objectives**

The primary purpose of this randomized study is to demonstrate that the 4GT Test lens senofilcon A with new UV-blocker, in its final lens design ECL600, meets the design validation requirements related to overall CLUE comfort, logMAR visual acuity, quality of vision in bright light, eye health, and fit acceptance.

## Secondary Objectives

The secondary objective of this study is to demonstrate that the Test lens is equal or better than marketed product senofilcon A (ACUVUE OASYS®, Johnson & Johnson Vision Care, Inc.) with regards to overall CLUE vision and handling.

Other observations of interest include adverse events, keratometry, surface characteristics (deposits and wettability), daily wear time, reasons for discontinuation, and lens damage.

# 2.2. Endpoints

# 2.2.1 Primary Efficacy Endpoints:

#### **CLUE Overall Comfort**

Overall comfort scores will be assessed using the Contact Lens User Experience (CLUE<sup>TM</sup>)<sup>7</sup> questionnaire at the two-week follow-up. CLUE is a validated patient-reported outcomes questionnaire to assess patient-experience attributes of soft, disposable contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE<sup>TM</sup> scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120. A 5-point increase in an average CLUE<sup>TM</sup> score translates into 10% shift in the distribution of scores for population of soft contact lens wearers.<sup>7</sup> The handling scores will be generated using the flexMIRT software Version 3 or higher (Chapel Hill, NC).

# Distance Monocular Contact Lens Visual Acuity

Distance monocular contact lens visual performance (logMAR) is assessed for each subject eye at the two-week follow-up evaluation using EDTRS charts using high illumination and high contrast charts.

# Vision Satisfaction in Bright Lighting

Vision satisfaction in bright lighting will be assessed using the individual item (Item ID: V015\_1) "I was satisfied with the quality of my vision in bright lighting" from the CLUE<sup>TM</sup> questionnaire. This item uses the response scale, 1: Strongly Disagree, 2: Disagree, 3: Neither Agree nor Disagree, 4: Agree and 5: Strongly Agree.

# 2.2.1. Primary Safety Endpoints:

## Slit Lamp Findings (Grade 3 or Higher)

Slit Lamp Findings will be assessed for each subject eye at all study visits (schedule and unscheduled). The percentage of eyes with Grade 3 or higher slit lamp findings will be analyzed and will include corneal infiltrates.

# Fit Acceptance Rate

Acceptable lens fit will be assessed at all study visits (scheduled and unscheduled) for each subject eye. Fit acceptance rate will be based on the lens fit acceptance of eyes wearing the Test lens only. Fit rates of the Control lens will also be collected but are not a primary endpoint.

# 2.2.2. Secondary Endpoints:

## **CLUE** Overall Vision and Handling

Overall vision and handling scores will be assessed using the Contact Lens User Experience (CLUE)<sup>7</sup> questionnaire at the two-week follow-up.

CR-6305, v4.0 Amendment 3.0 JJVCI CONFIDENTIAL

# 2.2.3. Other Endpoints:

# Average daily wear time (in Hours):

Average daily wear time will be calculated as the number of hours between subjects reported time of insertion and time of removal of the study lenses, on an average day, at 2-Week Follow-up evaluation.

# Subject's Reported Ocular Symptoms:

Frequency and severity by eye of subject's reported ocular symptoms and problems with the study lens at fitting and post-fitting evaluation visits including unscheduled visits.

Severity of the symptoms can be:

- 0 = Not Applicable or Not Recorded;
- 1 = Mild and results in little or no interference with lens wear;
- 2 = Moderate AND/OR occasionally interferes with lens wear;
- 3 = Severe AND/OR frequently interferes with lens wear.

The related procedure is explained in \_\_\_\_\_\_ of the study protocol.

# Lens fitting characteristics:

Frequency by eye of mechanical lens fitting characteristics at fitting and 2-Week Follow-up evaluations. Lens fitting characteristics to be reported are:

- Lens Centration Grade
- Decentered Direction
- Limbal Exposure Grade
- Edge Lift (Present or Absent)
- Primary Gaze Movement Grade
- Upgaze Movement Grade
- Lens Tightness Grade (Push-up Test)
- Acceptable Fitting (yes/no)

# Additional Endpoints

- Adverse events
- Discontinuation
- Reasons for discontinuation
- Unscheduled lens replacement
- Reasons for unscheduled lens replacement including lens damage.

## 2.3. Hypotheses

## 2.3.1. Primary Hypotheses

All the following primary hypotheses must be met for the objectives of this study to be satisfied:

1. Subjects wearing the JJVCI Investigational contact lenses on a daily wear basis will have patient reported comfort at the 2-Week Follow Up visit that is non-inferior to that of

- subjects wearing predicate device on a daily wear basis. A non-inferiority margin of -5 CLUE points will be used.
- 2. Subjects wearing the JJVCI Investigational contact lenses on a daily wear basis will report distance monocular visual acuity (logMAR: bright room luminance/high contrast charts) at the 2-Week Follow Up visit that is non-inferior to that of subjects wearing predicate device on a daily wear basis. A non-inferiority margin of 0.05 logMAR will be used.
- 3. Subjects wearing the JJVCI Investigational contact lenses on a daily wear basis will have patient reported outcome (Agree and Strongly Agree) on the Quality of Vision in Bright Light at the 2-Week Follow Up visit that is non-inferior to that of subjects wearing predicate device on a daily wear basis. A non-inferiority margin of 10% will be used.
- 4. Subjects wearing the JJVCI Investigational contact lenses on a daily wear basis will have a percentage of any Grade 3 or higher slit lamp findings at all visits (scheduled and unscheduled) that is non-inferior to that of subjects wearing predicate device on a daily wear basis. A non-inferiority margin of 5% will be used.
- 5. At least 90% of eyes wearing the JJVCI Investigational contact lenses on a daily wear basis will have acceptable fits across the fitting and follow-up visits.

# 2.3.2. Secondary Hypotheses

- 1. Subjects wearing the JJVCI Investigational contact lenses on a daily wear basis will have patient reported handling at the 2-Week Follow Up visit that is non-inferior to that of subjects wearing predicate device on a daily wear basis. A non-inferiority margin of -5 CLUE points will be used.
- 2. Subjects wearing the JJVCI Investigational contact lenses on a daily wear basis will have patient reported vision at the 2-Week Follow Up visit that is non-inferior to that of subjects wearing predicate device on a daily wear basis. A non-inferiority margin of -5 CLUE points will be used.

#### 3. TARGETED STUDY POPULATION

## 3.1. General Characteristics

Healthy adults of any race or ethnicity will be invited to participate. The eligible participants will be habitual wearers of spherical soft contact lenses as described below in Sections 3.2 and 3.3.

## 3.2. Inclusion Criteria

Potential subjects must satisfy all of the following criteria to be enrolled in the study:

# Inclusion Criteria after Screening

- 1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
- 2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
- 3. Between 18 and 49 (inclusive) years of age at the time of informed consent.
- 4. Eligible presbyopes will be those that wear full distance contact lenses in both eyes, then wear reading glasses over them when needed for near vision.
- 5. The subject is a current spherical soft contact lens wearer in both eyes with a minimum of 6 hours/day and 5 days/week wear time over the last 30 days by self-report.
- 6. Subjects must be able and willing to wear the study lenses at least 6 hours a day, a minimum of 5 days per week
- 7. Subjects must own a wearable pair of distance spectacles.

#### Inclusion Criteria after Baseline

- 8. The subject's vertex-corrected spherical equivalent distance refraction must be in the range of -1.00 to -6.00 D (inclusive) in each eye.
- 9. The subject's refractive cylinder must be 0.00 to -1.00 D (inclusive) in each eye.
- 10. The subject must have a spherocylindrical best corrected distance Snellen visual acuity of 20/25<sup>+3</sup> or better in each eye.

## 3.3. Exclusion Criteria

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

# Exclusion Criteria after Screening:

- 1. Currently pregnant or lactating (subjects who become pregnant during the study will be discontinued).
- 2. Any active or ongoing systemic disease (e.g., Sjögren's Syndrome), infectious disease (e.g., hepatitis, tuberculosis), contagious immunosuppressive diseases (e.g., HIV), autoimmune disease (e.g. rheumatoid arthritis).
- 3. Subjects taking suspect oral medications for less than one year. (See Section 3.3.1 for suspect medications and more details).
- 4. Any prescribed or over the counter (OTC) ocular medication.
- 5. Any known hypersensitivity or allergic reaction to Optifree® PureMoist® multi-purpose care solution or Eye-Cept® rewetting drop solution.
- 6. Toric, extended wear, monovision or multi-focal contact lens correction.
- 7. Any previous or planned (during the course of the study) ocular surgery (e.g., PRK, LASIK, etc.).
- 8. Participation in any contact lens or lens care product clinical trial within 30 days prior to study enrollment.

- 9. Participation in clinical trials involving the Test lens within 3 months prior to study enrollment.
- 10. Employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician).
- 11. Binocular vision abnormality or strabismus by self-report or prior medical history.
- 12. History of recurrent corneal erosions, herpetic keratitis, or pathological dry eye.

## Exclusion Criteria after Baseline

- 13. Any active ocular allergies, infections or other ocular abnormalities (entropion, extrusions, chalazia, recurrent styes, glaucoma) that the investigator determines may interfere with the outcomes of this study or otherwise contraindicate participation in the study.
- 14. Any Grade 2 or greater slit lamp findings (e.g., edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) on the FDA Slit Lamp Classification Scale.
- 15. Any previous history or signs of a contact lens-related corneal inflammatory event (e.g., past peripheral ulcer or round peripheral scar) within the past 3 years of otherwise successful contact lens wear.

# 3.3.1. Systemic Medications

Certain systemic medications are known to have a higher likelihood to interfere with contact lens wear, chiefly by disrupting the tear film. Several articles<sup>1,2,3</sup>, websites<sup>4,5</sup>, and text book chapters<sup>6,7</sup> discuss this topic with the general consensus shown in Table 1. Subjects taking these medications on a continual (year-round, routine) basis that have demonstrated successful contact lens wear for at least one year will generally be allowed to participate in this study. Subjects taking these medications on a routine basis but less than one year will not be allowed to participate in the study.

Note that subjects taking these medications on a temporary basis (e.g., antihistamines for seasonal allergy) will be allowed to participate if the medication has sufficient time to leave the body prior to the study. This is dependent on the half-life of the drug, body weight / fat, age, genetics, liver / kidney function, and metabolism of the subject. Given these unknowns, subjects taking the medications on a temporary basis must have ceased that medication at least one month prior to signing the informed consent.

<sup>&</sup>lt;sup>1</sup> Gomes, José Alvaro P., et al. "TFOS DEWS II iatrogenic report." The ocular surface 15.3 (2017): 511-538.

<sup>&</sup>lt;sup>2</sup> Silbert, Joel A. "A review of therapeutic agents and contact lens wear." Journal of the American Optometric Association 67.3 (1996): 165-172.

<sup>&</sup>lt;sup>3</sup> Muntingh, G. L. "Drug and contact lens interactions." South African Family Practice 47.8 (2005): 24-28.

<sup>&</sup>lt;sup>4</sup> https://www.clspectrum.com/issues/2003/september-2003/medication-effects-on-the-anterior-segment-and-con

<sup>&</sup>lt;sup>5</sup> http://www.richmondeye.com/ocular-side-effects-of-medications/

<sup>&</sup>lt;sup>6</sup> Lima, Claudia Assis, Newton Kara-Jose, and Jason J. Nichols. "Indications, Contraindications, and Selection of Contact Lenses." Contact Lenses in Ophthalmic Practice. Springer, New York, NY, 2004. 7-16.

<sup>&</sup>lt;sup>7</sup> Bartlett, Jimmy D., and Siret D. Jaanus. "Clinical ocular pharmacology." (2008): 575-578.

Table 1: Disallowed systemic medications (less than one year of continual use).

| Class of Drug | Common Indication(s) | Common Examples |
|---|---|---|
| Estrogens | Menopause, osteoporosis, vaginitis | Vagifem, Estrace, Climara,<br>Vivelle-Dot, Premarin, Minivelle,<br>etc., |
| Antihistamines | Allergic rhinitis, sedation, hives,<br>allergic conjunctivitis, skin allergy,<br>itching, motion sickness | Hydroxyzine, Promethegan,<br>Phenadoz, Vistaril, Claritin,<br>Zyrtec, Astepro, Astelin, Optivar,<br>Pataday, Allegra, Benadryl, etc., |
| Anticholinergics | Irritable bowel syndrome, Parkinson's disease, peptic ulcer, cystitis, nasal congestion, cold symptoms, overactive bladder, COPD | Bentyl, Spiriva, Atrovent,<br>Hyosyne, Levsin, Symax Fastab,<br>Symax SL, Homax SL, Cogentin,<br>Transderm Scop, etc., |
| Beta-blockers | Hypertension, angina, heart attack,<br>migraine, atrial fibrillation, adrenal<br>cancer, essential tumor, glaucoma | Toprol XL, Lopressor, Tenormin,<br>Propranolol, Timoptic, Trandate,<br>Inderal LA, etc., |
| Psychotropics | Antipsychotic (schizophrenia, mania), antidepression, antiobsessive, antianxiety, mood stabilizer, stimulants (ADHD) | Zoloft, Celexa, Prozac, Lexapro,<br>Effexor, Cymbalta, Ativan, Xanax,<br>Desyrel, Wellbutrin, etc., |
| Vitamin A<br>analogs | Cystic acne | Isotretinoin |

#### 3.4. Enrollment Strategy

Study subjects will be recruited from the Institution/clinical site's subject database and utilizing Institutional Review Board (IRB) approved materials.

#### 4. STUDY DESIGN AND RATIONALE

# 4.1. Description of Study Design

This study is a randomized, 2-visit, partially subject-masked, 2-arm parallel, dispensing trial. Approximately 236 subjects (118 subjects /arm) will be screened and enrolled to ensure that at least 224 subjects (112 subjects/arm) to complete.

The study begins with an initial visit (Visit 1). If a subject is found to meet all eligibility criteria, they will be randomized to one of two study lenses (Test or Control) in a bilateral fashion.

If the subject is dispensed study lenses at the initial visit, one follow-up visit will be conducted. The follow-up visit will occur approximately two weeks after the initial visit. Unscheduled follow-up visits may occur during the study. Subjects will be advised to wear the study lenses at least

five (5) days per week for at least six (6) hours per day for a period of two weeks. There is no planned lens replacement scheduled for during this study.

# 4.2. Study Design Rationale

The purpose of this study is to provide evidence that the investigational contact lens, senofilcon A with new-UV blocker meets all criteria specified by the Customer Requirements Document (CRD). Since this contact lens was approved for daily wear at a replacement rate of 2-weeks, a parallel study design with a 2-week follow-up evaluation was chosen as the most optimal design to evaluate the criteria specified in the CRD.

# 4.3. Enrollment Target and Study Duration

- Approximately 112 subjects are targeted to complete the Test arm of the study, and an additional 112 subjects are targeted to complete the Control arm of the study.
- 10 clinical sites will be recruited to participate, and each site will enroll approximately 20-24 subjects.
- Enrollment is defined at the point when the Informed Consent is signed. Termination is defined at the completion of the Final Evaluation.
- Each site will have approximately 2 weeks to enroll all their subjects unless otherwise approved by the Sponsor. Each subject will be in the study approximately 2 weeks, making the entire study approximately 4 weeks in duration.

**Table 2**: Target number of subjects by arm and site

| | Test | Control | Total |
|-------------------------|-------|---------|-------|
| Randomization | 116 | 116 | 232 |
| Completion | 112 | 112 | 224 |
| Number of sites | 10 | 10 | 10 |
| Subjects/site (Min-Max) | 10-12 | 10-12 | 20-24 |

## 5. TEST ARTICLE ALLOCATION AND MASKING

#### **5.1.** Test Article Allocation

A computer-generated randomization scheme will be used to randomly assign subjects, in blocks of 4, to one of the two possible study lenses (TEST or CONTROL). The random scheme will be generated using the PROC PLAN procedure from Statistical Analysis System (SAS) Software Version 9.4 or higher (SAS Institute, Cary, NC).

The study site must follow the randomization scheme provided and complete enrollment according to the randomization list and not pre-select or assign subjects. The randomized assignment of subjects will be performed at the first visit prior to the first fitting. The following must have occurred prior to randomization:

- Informed consent has been obtained
- Subject meets all the inclusion / not meets exclusion criteria
- Subject history and baseline information has been collected.

# 5.2. Masking

The dynamic nature of the Test lens makes it impossible to completely mask the study lens assignment. The subjects will be aware if they are wearing a photochromic lens or non-photochromic lens due to the function nature of the photochromic dye. Additionally, there is a slight difference in physical appearance between the Test and Control lenses when the Test lens is activated by outdoor light that makes it difficult to mask investigative personnel. However, the Control lens will be masked in the event that OASYS is the subject's habitual lens by chance, making this a partial-subject masked study.

Every attempt will be made to keep the other clinical trial personnel involved in the study (e.g. Data management, Biostatistician and Clinical Operations) unaware of the lens assignment. The identity of the study lenses will be masked by over labeling the blister packs with a label containing the study number, lot number, sphere power, expiration date and the randomization codes. Only the personnel involved in the over labeling and the Statistician generating the randomization scheme will have access to the decode information translating the randomization codes into Test and Control arms. The medical monitor will also have access to the decode information in case breaking the mask is necessary for the urgent medical treatment of a subject.

# 5.3. Procedures for Maintaining and Breaking the Masking

The test articles mask shall not be broken unless information concerning the lens type is necessary for the urgent medical treatment of a subject. The Sponsor must be notified before the mask is broken.

When dispensing test articles, the following steps should be followed to maintain randomization codes:

- 1. Investigator or designee (documented on the Delegation Log) will consult the lens fitting schedule/randomization scheme to obtain the test article assignment for that subject prior to dispensing
- 2. Investigator or designee will record the subject's number on the appropriate line of the randomization scheme
- 3. Investigator or designee will pull the appropriate test articles from the study supply. All test articles that are opened, whether dispensed (placed/fit on eye or dispensed outside the clinical site) or not, must be recorded on the Test Article Accountability Log in the "Dispensed" section

#### 6. STUDY INTERVENTION

# 6.1. Identity of Test Articles

The following contact lenses will be used in this study:

Table 3: Test Articles

| | Control | Test |
|---|---|---|
| Name | OASYS | ECL600 |
| Manufacturer | JJVCI | JJVCI |
| Lens Material | senofilcon A | senofilcon A |
| Nominal Base Curve @ 22°C | 8.4 | 8.4 |
| Nominal Diameter @ 22°C | 14.0 | 14.0 |
| Nominal Distance Powers (D) | -1.00 to -6.00 in 0.25 | -1.00 to -6.00 in 0.25 |
| 1 (20 45) | steps | steps |
| Water Content (%) | 38 | 38 |
| Center Thickness (-3.00 D) | 0.070 | 0.085 |
| Oxygen Permeability (Dk) | 103 | 103 |
| Modality in Current Study | Daily wear | Daily wear |
| Replacement Frequency | Single use | Single use |
| Packaging Form (vial, blister, etc.) | Sterile blister pack | Sterile blister pack |

There are 21 powers (sku's) from -1.00 through -6.00 D. Approximately 90 lenses per sku will be made available based on the following factors: sample size, bilateral wear, biweekly replacement, safety margin of 2x, and US distribution model.

# 6.2. Ancillary Supplies/Products

The following solutions will be used in this study:

Table 4: Ancillary Supplies

| | Solution 1 | Solution 2 |
|---|---|---|
| Solution Name /<br>Description | Opti-Free® PureMoist® | Eye-Cept®<br>Rewetting Drops |
| Lot Number or Other<br>Identifier | Varies | Varies |
| Manufacturer | Alcon Laboratories, Fort Worth, TX | Optics Laboratories |
| Maximum<br>Preservative | 0.001% polyquaternium-1, 0.0006% myristamidopropyl dimethylamine | NA |

## 6.3. Administration of Test Articles

Test articles will be dispensed to subject meeting all eligibility requirements, including any dispensing requirements set forth in this clinical protocol. Subjects will be dispensed an adequate supply of test articles to complete the study. Lost or damaged test articles may be replaced at the discretion of the Investigator and/or the Sponsor.

# 6.4. Packaging and Labeling

The Control articles will be packaged in their commercial blister packs with investigational overlabel to mask their identity. The Test articles will be packaged in blisters as the primary packaging and labeled with investigational foil. The test articles will be in plastic bags as the secondary packaging form. The sample study label is shown below:





# 6.5. Storage Conditions

Test articles will be maintained at ambient temperatures at the clinical site. Test articles must be kept under secure conditions and out of direct sunlight.

## 6.6. Collection and Storage of Samples

All worn study lenses will be collected from the subject, placed in labeled glass vials with Opti-Free® PureMoist®, and stored refrigerated or frozen until they are shipped back to the Sponsor. The lenses will be shipped in special containers to keep the lenses refrigerated.

When possible, any lens or test article associated with an Adverse Events and/or a Product Quality Complaint must be retained and stored in a glass vial with moderate solution pending directions from the sponsor for potential return back to JJVCI.

# 6.7. Accountability of Test Articles

JJVCI will provide the Investigator with sufficient quantities of study articles and supplies to complete the investigation. The Investigator is asked to retain all lens shipment documentation for the test article accountability records.

Test article must be kept in a locked storage cabinet, accessible only to those assigned by the Investigator for dispensing. The Investigator may delegate this activity to authorized study site personnel listed on the Site Delegation Log. All test articles must be accounted. This includes:

- 1. What was dispensed for the subject for trial fitting, to wear out of the office, or issued for the subject to replace appropriately between visits
- 2. What was returned to the Investigator unused
- 3. The number and reason for unplanned replacements

Following final reconciliation of test articles by the monitor, the Investigator or monitor will return all unused test articles to JJVCI.

If there is a discrepancy between the shipment documents and the contents, contact the study monitor immediately.

## 7. STUDY EVALUATIONS

# 7.1. Time and Event Schedule

Table 5: Time and Events

| Visit Information | Visit 1 | Visit 2 |
|---|---|---|
| | Screening, Baseline, | Follow-up, |
| | Treatment 1 | Final Evaluation |
| Time Point | Day 1 | Day 14 ± 1 |
| Estimated Visit Duration | 2.5 hours | 1.5 hours |
| Statement of Informed Consent | X | |
| Demographics | X | |
| Medical History/Concomitant Medications | X | X |
| Habitual Contact Lens Information | X | |
| Inclusion/Exclusion Criteria | X | |
| Baseline Questionnaires | X | |
| Entrance Visual Acuity | X | |
| Iris Color | X | |
| Keratometry | X | X |
| Subjective Sphero-Cylindrical Refraction | X | X |
| Slit Lamp Biomicroscopy | X | X |
| Lens Selection | X | |
| Lens Insertion & Settling | X | |
| Visual Acuity and Over Refraction | X | |
| Lens Power Modification | X | |
| Subject Reported Ocular Symptoms | X | X |
| Visual acuity (distance Snellen) | X | X |
| Lens Fit Assessment | X | X |
| Lens Wettability | X | X |
| Dispense Patient Instruction Guide | X | |
| Dispense Test Article | X | |

| Visit Information | Visit 1 | Visit 2 |
|---|---|---|
| | Screening, Baseline, | Follow-up, |
| | Treatment 1 | Final Evaluation |
| Time Point | Day 1 | Day 14 ± 1 |
| Estimated Visit Duration | 2.5 hours | 1.5 hours |
| Lens wear Compliance | | X |
| Wearing Time and Compliance | | X |
| Follow-up Questionnaire | | X |
| Distance ETDRS logMAR Visual Acuity | | X |
| Surface Deposits | | X |
| Study Completion | | X |
| Lens Removal and Storage | | X |
| Final Evaluation | | X |

# 7.2. Detailed Study Procedures

Range and Article and the Commission of March 2012 and the Commiss

VISIT 1

The subjects must present to Visit 1 wearing their habitual contact lenses.

| | Visit 1: Screening | | |
|---|---|---|---|
| Step | Procedure | Details | |
| 1.1 | Statement of<br>Informed Consent | Each subject must read, understand, and sign the Statement of Informed Consent before being enrolled into the study. The Principal Investigator or his/her designee conducting the informed consent discussion must also sign the consent form. Note: The subject must be provided a signed | |
| r. | | copy of this document. | 3 |
| 1.2 | Demographics | Record the subject's date of birth, gender, race and ethnicity. | |
| 1.3 | Medical History and<br>Concomitant<br>Medications | Questions regarding the subjects' medical history and concomitant medications. | |
| 1.4 | Habitual Lenses | Questions regarding the subject's habitual lens type and parameters. | |
| 1.5 | Eligibility after<br>Screening | All responses to Screening Inclusion Criteria questions must be answered "yes" and all responses to Exclusion Criteria must be answered "no" for the subject to be considered eligible. | |

| 1 | Visit 1: Screening | |
|---|---|---|
| Step | Procedure | Details |
| | | If the subject is deemed to be ineligible after screening, proceed to Final Evaluation and complete Subject Disposition. Refraction and Biomicroscopy forms are not required. |

| | Visit 1: Baseline | |
|---|---|---|
| Step | Procedure | Details |
| 1.6 | Baseline<br>Questionnaire | The subject will respond to the CLUE Baseline Questionnaire. |
| 1.7 | Entrance Visual<br>Acuity | Record the distance Snellen visual acuity (OD, OS, and OU) to the nearest letter with their habitual contact lens correction in place. Subjects must read the smallest line until at least 50% of the letters are read incorrectly. |
| 1.8 | Remove Habitual<br>Lens | The subject's habitual lenses will be removed and stored in their own lens case. If they forgot to bring their lens case, one will be provided to them. |
| 1.9 | Iris Color | The investigator will record the subject's iris color based on the scale provided. |
| 1.10 | Keratometry | Record the keratometry readings OD and OS in diopters. This can come from any appropriate instrument so long as the same instrument is used at the Final Evaluation. |
| 1.11 | Subjective Sphero-<br>cylindrical Refraction | Complete subjective spherocylindrical refraction and record the resultant distance visual acuity (OD, OS, and OU) to the nearest letter. Best corrected distance visual acuity (BVA) must be 20/25+3 or better in each eye. |
| 1.12 | Slit Lamp<br>Biomicroscopy | FDA Slit Lamp Classification Scale will be used to grade the findings and determine eligibility. If any of these slit lamp findings are grade 2 or higher, the subject may not continue at this time, but may return up to one additional time to determine eligibility. If after a total of 2 attempts the subject is deemed |

| | Visit 1: Baseline | |
|---|---|---|
| Step | Procedure | Details |
| | | ineligible, then complete the Final Evaluation. If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops or saline may be instilled. |
| 1.13 | Eligibility after<br>Baseline | All responses to Inclusion Criteria questions must be answered "yes" and all responses to Exclusion Criteria questions must be answered "no" for the subject to be considered eligible. If subject is deemed to be ineligible after the first or second baseline, proceed to Final Evaluation and complete all forms. |

| | Visit 1: Treatment 1 Lens Fitting | |
|---|---|---|
| Step | Procedure | Details |
| 1.14 | Lens Selection | Assign the study lens based on the randomization scheme. Select the contact lens power based on subjective refraction. Record the test condition. |
| 1.15 | Lens Insertion | The Investigator or the subject inserts the study lenses. Record the time of lens insertion. Check for lens damage under the slit lamp before proceeding with lens settling. Replace damaged lenses if applicable. |
| 1.16 | Lens Settling | Allow the study lenses to settle for a minimum of 5 minutes. |
| 1.17 | Subjective Best<br>Sphere Over<br>Refraction | Perform subjective best sphere refraction over the study lenses with a phoropter (adopt the maximum plus to maximum visual acuity (MPMVA) approach and use the duo-chrome, binocular blur, or other suitable test for binocular balancing) and record the best corrected distance Snellen visual acuity to the nearest letter (OD, OS, and OU). |

| 5 | Visit 1: Treatment 1 Lens Fitting | | |
|---|---|---|---|
| Step | Procedure | Details | |
| 1.18 | Lens Power<br>Modification (if<br>applicable) | Adjust the lens power if the subject's best sphere over-refraction is not plano. For each power modification, repeat steps (1.15-1.17). One power modification is allowed per eye. | |
| 1.19 | Time Interval | Please wait for at least 10 minutes from final lens insertion to continue. | |
| 1.20 | Subject Reported<br>Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire. | |
| 1.21 | Visual Acuity | Record the distance Snellen visual acuity with<br>the contact lenses (OD, OS, and OU) to the<br>nearest letter. Smaller lines must be shown until<br>the subject incorrectly identifies at least 50% of<br>the letters. | |
| 1.22 | Subjective Lens Fit<br>Assessment | Evaluate overall lens fit acceptance (acceptable or unacceptable) based on centration, movement and other fitting characteristics. An unacceptable fit is deemed by one of the following criteria: Imbal exposure at primary gaze or with extreme eye movement edge lift excessive movement in primary and up gaze insufficient movement in all three of the following conditions: primary gaze, up gaze, and Josephson push up Note: if lens fit is unacceptable subject will be discontinued from the study. | |
| 1.23 | Lens Wettability | Perform the white light lens wettability procedure and record the results. | P |
| 1.24 | Continuance | For the subject to continue in the study, they must meet all three of the following criteria: • Visual acuity is 20/30 or better OD and OS • The lens fit is acceptable OD and OS • Investigator approval. | |

| 5: | Visit 1: Treatment 1 Lens Fitting | |
|---|---|---|
| Step | Procedure | Details |
| | | If the Investigator does not approve the dispensing of the first study lens based on subject feedback (e.g., unsatisfactory comfort), then the study is terminated for that subject. |
| 1.25 | Dispense | <ol> <li>The lenses will be dispensed for 13-15 days</li> <li>The subjects should wear their lenses similar to the inclusion criteria: ≥ 6 hours per day, ≥ 5 days per week.</li> <li>The lenses will be worn as daily wear only.</li> <li>All subjects will be provided Opti-Free PureMoist to be used in a rub regime.</li> <li>Preservative-free rewetting drops are permitted if needed.</li> <li>A patient instruction booklet will be provided.</li> <li>The lenses must be stored in the supplied case out of direct sunlight.</li> <li>Note 1: In the event a lens is lost or damaged, the subject will return to the investigator site for replacement (extra lenses cannot be given at the dispensing visit).</li> <li>Note 2: The subject's habitual contact lenses cannot be worn at any time during the study.</li> <li>Note 3: Instruct subjects to bring their spectacles to the next visit.</li> </ol> |

# VISIT 2

The follow-up will occur 13-15 days following Visit 1. The subjects must enter the visit wearing their study contact lenses.

| | Visit 2: Treatment 1 Follow-Up 1 | | |
|---|---|---|---|
| Step | Procedure | Details | |
| 2.1. | Adverse Events and<br>Concomitant<br>Medications Review | Review any changes to the subject's medical history or concomitant medications from the previous study visit. Record any changes, and any adverse events. | |
| 2.2. | Wearing Time | Record the average wearing time and comfortable wearing time. | r. |
| 2.3. | Compliance | Confirm compliance with the prescribed wear schedule. | |
| 2.4. | Subject Reported<br>Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire. | |
| 2.5. | Follow-Up<br>Questionnaires | The subject will respond to the Follow-Up Questionnaires. | |
| 2.6. | Visual Acuity | Record the distance Snellen visual acuity with<br>the contact lenses (OD, OS, and OU) to the<br>nearest letter. Subjects must read the smallest<br>line until at least 50% of the letters are read<br>incorrectly. | |
| 2.7. | Distance ETDRS LogMAR Visual Acuity | Perform 4 m distance ETDRS LogMAR visual acuity test OD and OS under the following conditions: Bright room illumination / high contrast charts a. Room illumination > 400 lux b. Chart luminance 120-200 cd/m² c. One high contrast chart per eye. 1) OD: chart HC-1 2) OS: chart HC-2 | |
| 2.8. | Subjective Lens Fit<br>Assessment | Evaluate overall lens fit acceptance (acceptable or unacceptable) based on centration, movement and other fitting characteristics. An unacceptable fit is deemed by one of the following criteria: Imbal exposure at primary gaze or with extreme eye movement edge lift | |

| Visit 2: Treatment 1 Follow-Up 1 | | |
|---|---|---|
| Step | Procedure | Details |
| | | <ul> <li>insufficient or excessive movement in<br/>all three of the following conditions:<br/>primary gaze, up gaze, and Josephson<br/>push up</li> </ul> |
| 2.9. | Lens Wettability | Perform the white light lens wettability procedure and record the results. |
| 2.10. | Surface Deposits | Record any front and back surface lens deposits. |
| 2.11. | Lens Removal & Storage | Both lenses will be removed and stored wet in a labeled container with Opti-Free PureMoist. The lenses can be stored refrigerated or frozen prior to shipment back to the Sponsor. Lenses will be stored at JJVCI for 45 days after LSLV for laboratory testing (Section 7.4). |
| 2.12. | Slit Lamp<br>Biomicroscopy | FDA Slit Lamp Classification Scale will be used to grade the findings. If the subject has a Grade 3 or higher slit lamp finding, it will be recorded as an Adverse Event and the subject will be followed to resolution. Adverse events must be reported to the JJVCI monitors immediately. If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops may be instilled. |

# FINAL EVALUATION

The final evaluation will ordinarily take place immediately following the last scheduled follow-up visit per the study protocol. It may also take place at any point the subject discontinues the study or is terminated from the study.

| | Final Evaluation | |
|---|---|---|
| Step | Procedure | Details |
| F.1 | Final Exam Form | Indicate if the subject completed the study successfully. If subject discontinued from the study, indicate the reason. |
| F.2 | Keratometry | Record the keratometry readings OD and OS in diopters. This can come from any appropriate instrument so long as the same instrument was used at the Baseline Evaluation. |

| Final Evaluation | | |
|---|---|---|
| Step | Procedure | Details |
| F.3 | Subjective<br>spherocylindrical<br>Refraction | Perform bare-eye subjective spherocylindrical refraction with a phoropter and record the best corrected <u>distance</u> visual acuity to the nearest letter (OD, OS, and OU). |

## 7.3. Unscheduled Visits

If, during the investigation a symptomatic subject requires an unscheduled visit to the clinical site, the following information will be collected at a minimum (if applicable):

- Chief complaint prompting the visit. If the reason is an adverse event, the applicable eCRF for the adverse event must be completed and subject record completed as appropriate
- Date and time of the visit and all procedures completed at the unscheduled visit
- · Review of adverse event and concomitant medications
- Documentation of any test article dispensed or collected from the subject, if applicable
- Slit lamp findings (using the Slit Lamp Classification Scale)

If the Investigator withdraws a subject from the study, the final study visit case report forms must be completed indicating the reason(s) why the subject was withdrawn. The subject record must be completed documenting the date and primary reason for withdrawal and the study CRA notified.

Any ocular and non-ocular Adverse Events that are ongoing at the time of the study visit will be followed by the Investigator, within licensure, until they have resolved, returned to pre-treatment status, stabilized, or been satisfactorily explained. If further treatment i.e., beyond licensure is required, the subject will be referred to the appropriate health care provider.

The following information will be collected during an unscheduled visit. The investigational sites only need to complete steps U.1, U.2, and U.6 for asymptomatic subjects that simply require a replacement lens.

| Unscheduled Visit | | | | | | |
|---|---|---|--|--|--|--|
| Step | Procedure | Details | | | | |
| U.1 | Chief Complaints | Record the subject's chief complaints for reasons for the unscheduled visit. | | | | |
| U.2 | Adverse Events and<br>Concomitant<br>Medications Review | Review any changes to the subject's medical history or concomitant medications from the previous study visit. Record any changes, and any adverse events. | | | | |
| U.3 | Entrance VA | Record the entrance distance visual acuity (OD, OS and OU) to the nearest letter. | | | | |
| Unscheduled Visit | | | | |
|---|---|---|--|--|
| Step | Procedure | Details | | |
| U.4 | Subjective Sphero-<br>cylindrical Refraction | The investigator will complete a subjective refraction (sphere and cylinder) and record the resultant distance visual acuity OD, OS, and OU to the nearest letter. | | |
| U.5 | Slit Lamp<br>Biomicroscopy | FDA Slit Lamp Classification Scale will be used to grade the findings. If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops may be instilled. | | |
| U.6 | Dispensing (if applicable) | Additional lenses may be dispensed if one is lost or torn during the wearing period. | | |
| U.7 | Exit Visual Acuity | Record the subject's exit distance visual acuity (OD, OS, and OU) to the nearest letter. | | |

## 7.4. Laboratory Procedures

The optical bench will be used to measure the light transmission characteristics for all worn Test lenses. The findings are for internal information only and will not be part of the final report.

#### 8. SUBJECTS COMPLETION/WITHDRAWAL

# 8.1. Completion Criteria

Subjects are considered to have completed the study if they:

- provided informed consent
- they are eligible
- Completed all required study visits

## 8.2. Withdrawal/Discontinuation from the Study

A subject will be withdrawn from the study for any of the following reasons:

- Subject death during the study period
- Subject withdrawal of consent
- Subject not compliant to protocol
- Subject lost to follow-up
- Subject no longer meets eligibility criteria (e.g. the subject becomes pregnant)
- Subject develops significant or serious adverse events causing discontinuation of study lens
  wear
- Subjects who have experienced a Corneal Infiltrative Event (CIE)
- Investigator's clinical judgment regarding the subject safety reasons (that it is in the best interest of the subject to stop treatment)
- · Subject missed a scheduled study visit

- Subject not compliant with study lens wear schedule
- Subject not successfully dispensed due to lack of efficacy and safety including poor vision, poor comfort or unacceptable fit
- Subject out of visit window visit with two or more days

For discontinued subjects, the Investigator will:

- Complete the current visit (scheduled or unscheduled)
- Complete the Final Evaluation, indicating the reason that the subject was discontinued from the study
- Record the spherocylindrical refraction with best corrected distance visual acuity
- Collect used test article(s) (worn or brought to the visit) from the subject
- Collect all unused test article(s) from the subject

An additional subject will be enrolled if a subject discontinues from the study prematurely.

In cases where a subject is lost to follow-up, every possible effort must be made to contact the subject and determine the reason for discontinuation/withdrawal. The measures taken to follow up must be documented including two written attempts and a certified letter (or equivalent) as the final attempt.

# 9. PRE-STUDY AND CONCOMITANT INTERVENTION/MEDICATION

Concomitant medications will be documented during screening and updated during the study. Suspect disallowed oral medications taken for less than one year on a continual (year-round, routine) basis are listed in Section 3.3.1. Document any prescribed or over the counter (OTC) ocular medication currently being taken.

#### 10. DEVIATIONS FROM THE PROTOCOL

Investigator will notify study sponsor upon identification of a protocol deviation. Major protocol deviations must be reported to the sponsor within 24 hours after discovery of the protocol deviation. The Investigator will report deviations per IRB/IEC requirements. All deviations will be tracked and corrective actions implemented as appropriate.

If it becomes necessary for the Investigator to implement a deviation in order to eliminate an immediate hazard to the trial subject, the Investigator may implement the deviation immediately without notification to the sponsor. Within 24 hours after the implemented deviation, the Investigator must notify and provide the rationale to the Sponsor and, as required, the IEC/IRB.

## 11. STUDY TERMINATION

The occurrence of one or more Unanticipated Serious Adverse Device Effect (USADE), or any SAE where the relationship to study agent cannot be ruled out, may result in stopping further dispensing of test article. In the event of a USADE or SAE, the Sponsor may unmask the treatment

CR-6305, v4.0 Amendment 3.0


regimen for the subject(s) and will discuss this with the Investigator before any further subjects are enrolled.

The Sponsor will determine when a study will be stopped. The Principal Investigator always has the discretion to initiate stopping the study based on patient safety or if information indicates the study's results are compromised.

JJVCI reserves the right to terminate the study at any time for any reason. Additionally, the IEC/IRB reserves the right to terminate the study if an unreasonable risk is determined. The study can be terminated by the Principal Investigator at the individual clinical site due to specific clinical observations, if in their opinion, after a discussion with JJVCI, it is determined that it would be unwise to continue at the clinical site.

JJVCI (and the IEC/IRB and DMC, if applicable) will evaluate all adverse events. If it is determined that an adverse event presents an unreasonable risk, the investigation, or that part of the investigation presenting the risk, will be terminated, as soon as possible.

Should the study be terminated (either prematurely or as scheduled), the Investigator will notify the IEC/IRB and Regulatory Authority as required by local regulatory requirements.

# 12. PROCEDURE FOR HANDLING PRODUCT QUALITY COMPLAINTS

A Product Quality Complaint (PQC) refers to any written, electronic, or oral communication that alleges deficiencies related to the identity, quality, durability, reliability, safety, effectiveness or performance of test articles after they have been released for clinical trial use.

Potential complaints may come from a variety of sources including but not limited to subjects, clinical research associates (CRA), clinical operations managers (COM), medical monitors, and site personnel, etc. The following are not considered product quality complaints:

- Subject satisfaction inquiries reported via "Subjective Questionnaires" and "Patient Reported Outcomes (PRO)"
- Clinical test articles that are stored improperly or damaged after receipt at the investigational site
- Lens replacements that occur due to drops/fall-outs
- Damage deemed by clinicians or clinical staff to be caused by handling by the user, and not indicative of a quality deficiency (i.e. tears, rips, etc.), only in situations where there is no deficiency alleged by the subject

Within 24 hours of site personnel becoming aware that a PQC has occurred, the PQC must be recorded in the EDC system, which will trigger an automatic email notification to the appropriate COM/CRA and Clinical QA representative. In cases where the EDC system in use is not configured to send automatic notifications or when an EDC system is not used, the COM/CRA is responsible for notifying Clinical QA upon discovery that a PQC has occurred.

Upon receipt of the EDC notification, the COM/CRA will contact the study site to collect additional information which will include:

- Date the complaint was received/recorded in the EDC System (Date of Sponsor Awareness)
- Who received the complaint
- Study number
- Clinical site information (contact name, site ID, telephone number)
- Lot number(s)
- Unique Subject Identifier(s)
- Indication of who first observed complaint (site personnel or subject)
- OD/OS indication, along with whether the lens was inserted
- Any related AE number if applicable
- Detailed complaint description (scheduled/unscheduled visit, wear time, symptoms, resolution of symptoms, etc.)
- Eye Care Provider objective (slit lamp) findings if applicable
- Confirmation of product availability for return (and tracking information, if available), or rationale if product is not available for return

Once a complaint is received, it will be assessed by the COM, CRA, or trained site personnel to determine if it is an Adverse Event/Serious Adverse Event (AE/SAE). If the complaint results in an AE/SAE, the COM/CRA, or trained site personnel will follow Section 13 of this protocol. If the AE/SAE was potentially the result of a product quality related deficiency, these procedures also applies and will be executed in parallel.

In some cases, a PQC form may be generated in EDC by the site in error. In this event, the PQC forms will be marked "Intentionally Left Blank" or "ILB". Justification for ILB must be documented.

#### 13. ADVERSE EVENTS

#### 13.1. Definitions and Classifications

**Adverse Event (AE)** – An AE is "any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the investigational medical device.

*Note 1* to entry: This definition includes events related to the investigational medical device or the comparator.

*Note 2* to entry: This definition includes events related to the procedures involved.

*Note 3* to entry: For users or other persons, this definition is restricted to events related to investigational medical devices."<sup>1</sup>

An AE includes any condition (including a pre-existing condition) that:

1. Was not present prior to the study, but appeared or reappeared following initiation of the study

- 2. Was present prior to the study, but worsened during the study. This would include any condition resulting from concomitant illnesses, reactions to concomitant medications, or progression of disease states
- 3. Pregnancy must be documented as an adverse event and must be reported to the clinical monitor and to the Sponsor immediately upon learning of the event

Serious Adverse Event (SAE) – An SAE is any untoward medical occurrence that:

- Results in death
- Is life threatening
- Requires in-patient hospitalization or prolongation of existing hospitalization
- Results in persistent or significant disability/incapacity (e.g., a sight threatening event, a significant persistent or permanent change, impairment, damage, or disruption to the subject's body)
- Is a congenital anomaly/birth defect, or
- Requires intervention to prevent permanent damage (the use of the test article resulting in
  a condition which requires medical or surgical intervention to preclude permanent
  impairment of the body structure or a body function). Important medical events that may
  not result in death, be life-threatening, or require hospitalization may be considered an SAE
  when, based upon appropriate medical judgment, they may jeopardize the patient or subject
  and may require medical or surgical intervention to prevent one of the outcomes listed in
  the above definition

Diagnoses and conditions that are considered Ocular Serious Adverse Events include, but not limited to:

- Microbial Keratitis (MK)
- Iritis (including cells in the anterior chamber)
- Permanent decrease in best spectacle corrected visual acuity equivalent to 2 acuity lines or greater
- Central Corneal Opacity
- Central Corneal Neovascularization
- Uveitis
- Endophthalmitis
- Hypopyon
- Hyphemia
- Penetration of Bowman's Membrane
- Persistent Epithelial Defect
- Limbal cell Damage leading to Conjunctivalization

**Significant Adverse Events** – Those events that are usually symptomatic and warrant discontinuation (temporary or permanent) of the test article (excluding Serious Adverse Events).

Diagnoses and conditions that are considered Ocular Significant Adverse Events include, but not limited to the following:

- Contact Lens Induced Peripheral Ulcer (CLPU)
- Significant Infiltrative Events (SIE)

- Superior Epithelial Arcuate Lesions (SEALs)
- Any Temporary Loss of >2 Lines of BSCVA
- Other grade 3 or higher corneal findings, such as abrasions or edema
- Non-contact lens related corneal events e.g. Epidemic Keratoconjunctivitis (EKC)
- Asymptomatic Corneal Scar
- Any corneal event which necessitates temporary lens discontinuation >2 weeks

**Non-Significant Adverse Events** – Those conditions that are usually asymptomatic and usually do not warrant discontinuation (temporary or permanent) of the test article. However, the Investigator may choose to treat as a precautionary measure.

Diagnoses and conditions that are considered Ocular Non-Significant Adverse Events include, but not limited to the following:

- Non-significant Infiltrative Event (NSIE)
- Contact Lens Papillary Conjunctivitis (CLPC)
- Superficial Punctate Keratitis (SPK)
- Conjunctivitis: Bacterial, Viral, Allergic
- Blepharitis
- Meibomianitis
- Contact Dermatitis
- Localized Allergic Reactions
- Any corneal event not explicitly defined as serious or significant adverse event, which necessitates temporary lens discontinuation <2 weeks

**Adverse Device Effect (ADE)** – An ADE is an "adverse event related to the use of an investigational medical device.

*Note 1* to entry: This definition includes adverse events resulting from insufficient or inadequate instructions for use, deployment, implantation, installation, or operation, or any malfunction of the investigational medical device.

*Note 2* to entry: This definition includes any event resulting from use error or from intentional misuse of the investigational medical device."

Unanticipated Adverse Device Effect (UADE) – Any serious adverse effect on health or safety or any life-threatening problem or death caused by, or associated with, the test article, if that effect, problem, or death was not previously identified in nature, severity, or degree of incidence in the investigational plan, Investigator's Brochure or protocol, or any other unanticipated serious problem associated with the test article that relates to the rights, safety and welfare of subjects.

#### 13.2. Assessing Adverse Events

In conjunction with the medical monitor, the Investigator will evaluate adverse events to ensure the events are categorized correctly. Elements of categorization will include:

- Seriousness/Classifications (see definition in Section 13.1)
- Causality or Relatedness i.e. the relationship between the test article, study treatment or study procedures and the adverse event (not related; unlikely related; possibly related; related see definition in Section 13.2.1)

- Adverse Event Severity Adverse event severity is used to assess the degree of intensity of the adverse event (mild; moderate; severe for all events see definition in Section 13.2.2)
- Outcome not recovered or not resolved; recovering or resolving; recovered or resolved with sequelae; recovered or resolved; death related to adverse event; unknown
- Actions Taken none; temporarily discontinued; permanently discontinued; other

## 13.2.1. Causality Assessment

**Causality Assessment** – A determination of the relationship between an adverse event and the test article. The test article relationship for each adverse event should be determined by the investigator using these explanations:

- Not Related- An adverse event that is not related to the use of the test article, study treatment or study procedures
- Unlikely Related An adverse event for which an alternative explanation is more likely, e.g. concomitant treatment, concomitant disease(s), or the relationship of time suggests that a causal relationship is not likely
- Possibly Related An adverse event that might be due to the use of the test article, or to the study treatment or study procedures. An alternative explanation, e.g. concomitant treatment, concomitant disease(s), is inconclusive. The relationship in time is reasonable. Therefore, the causal relationship cannot be excluded
- Related An adverse event that is listed as a possible adverse effect (device) or adverse reaction (drug) and cannot be reasonably explained by an alternative explanation, e.g. concomitant treatment of concomitant disease(s). The relationship in time is very suggestive, e.g. it is confirmed by de-challenge and re-challenge

# 13.2.2. Severity Assessment

**Severity Assessment** – A qualitative assessment of the degree of intensity of an adverse event as determined by the Investigator or reported to him/her by the subject. The assessment of severity is made irrespective of test article, study treatment or study procedure relationship or seriousness of the event and should be evaluated according to the following scale:

- Mild Event is noticeable to the subject, but is easily tolerated and does not interfere with the subject's daily activities
- Moderate Event is bothersome, possible requiring additional therapy, and may interfere with the subject's daily activities
- Severe Event is intolerable, necessitates additional therapy or alteration of therapy and interferes with the subject's daily activities

#### 13.3. Documentation and Follow-Up of Adverse Events

The recording and documenting of adverse events (ocular and non-ocular) begins when the subjects are exposed to the test article, study treatment or study procedure. Adverse events reported before the use of test article, start of study treatment, or study procedures will be recorded as medical history. However, if the condition deteriorates at any time during the study it will be recorded and reported as an AE. Untoward medical events reported after the subject's exit from the study will be recorded as adverse events at the discretion of the Investigator.

Upon finding an adverse event, the Principal Investigator will document the condition in the subject record and in the eCRFs. He/she will complete the Adverse Event /eCRF.

Complete descriptions of all adverse events must be available in the subject record. All Adverse Events including local and systemic reactions not meeting the criteria for "serious adverse events" shall be captured on the appropriate case report form or electronic data system. All adverse events occurring while the subject is enrolled in the study must be documented appropriately regardless of relationship.

It is the Investigator's responsibility to maintain documentation of each reported adverse event. All adverse events will be followed in accordance with applicable licensing requirements. Such documentation will include the following:

- Adverse event (diagnosis not symptom)
- Drawings or photographs (where appropriate) that detail the finding (e.g., size, location, and depth, etc.)
- Date the clinical site was notified
- Date and time of onset
- Date and time of resolution
- Adverse event classification, severity, and relationship to test articles, as applicable
- Treatment regimen instituted, including concomitant medications prescribed, in accordance with applicable licensing requirements
- Any referral to another health care provider if needed
- Outcome, ocular damage (if any)
- Likely etiology
- Best corrected visual acuity at the discovery of the event and upon conclusion of the event

In addition, if an infiltrate(s) is present, he/she will complete the Corneal Infiltrate Assessment eCRF. Where necessary, a culture of the corneal lesion will be collected to determine if the infection is microbial in nature. If cultures are collected, the date of culture collection and laboratory utilized will be recorded.

Changes in the severity of an AE shall be documented to allow an assessment of the duration of the event at each level of intensity to be performed. Adverse events characterized as intermittent require documentation of the onset and duration of each episode. Changes in the assessment of relationship to the Test Article shall also be clearly documented.

Subjects who present with an adverse event shall be followed by the Investigator, within licensure, until all signs and symptoms have returned to pre-treatment status, stabilized, or been satisfactorily resolved. If further treatment beyond licensure is required, the patient will be referred to the appropriate health care provider. The Investigator will use his/her clinical judgment as to whether a subject reporting with an adverse event will continue in the study. If a subject is discontinued from the study, it will be the responsibility of the Investigator to record the reason for discontinuation. The Investigator will also document the adverse event appropriately and complete the Adverse Event eCRF. Any subjects with ongoing adverse events related to the test article, study treatment or study procedures, as of the final study visit date, should be followed to

resolution of the adverse event or until referral to an appropriate health care provider, as recommended by the Investigator. Non-ocular adverse events that are not related to the test article, study treatment, or study procedures may be recorded as "ongoing" without further follow-up.

# 13.4. Reporting Adverse Events

The Investigator will notify the Sponsor of an adverse event by e-mail, facsimile, or telephone as soon as possible and no later than 24 hours from discovery for any serious /significant adverse events, and 2 days from discovery for any non-significant adverse event. In addition, a written report will be submitted by the Principal Investigator to the IEC/IRB according to their requirements (Section 13.4.2). The report will comment whether the adverse event was considered to be related to the test article, study treatment or study procedures.

# 13.4.1. Reporting Adverse Events to Sponsor

# **Serious/Significant Adverse Events**

The Investigator will inform the sponsor of all serious/significant adverse events occurring during the study period as soon as possible by e-mail, fax, or telephone, but no later than 24 hours following discovery of the event. The Investigator is obligated to pursue and obtain information requested by the Sponsor in addition to that information reported on the eCRF. All subjects experiencing a serious/significant adverse event must be followed up and all outcomes must be reported.

When medically necessary, the Investigator may break the randomization code to determine the identity of the treatment that the subject received. The Sponsor and study monitor should be notified prior to unmasking the test articles.

In the event of a serious/significant adverse event, the Investigator must:

- Notify the Sponsor immediately
- Obtain and maintain in the subject's records all pertinent medical information and medical judgment for colleagues who assisted in the treatment and follow-up of the subject
- Provide the Sponsor with a complete case history which includes a statement as to whether the event was or was not related to the use of the test article
- Notify the IEC/IRB as required by the IEC/IRB reporting procedure according to national regulations

# **Unanticipated (Serious) Adverse Device Effect (UADE)**

In the event of an Unanticipated (Serious) Adverse Device Effect (UADE), the Investigator will submit a report of the UADE to the Sponsor and IEC/IRB as soon as possible, but no later than 24 hours after the Investigator first learns of the effect. This report is in addition to the immediate notification mentioned above.

The Sponsor must conduct an evaluation of the UADE and must report the results of the evaluation to FDA, the IEC/IRB and participating Investigators within 10 working days after the Sponsor first receives notification of the effect.

#### **Non-Serious Adverse Events**

All non-serious adverse events, including non-serious adverse device effects, will be reported to the sponsor by the Investigator no later than 2 days from discovery.

## 13.4.2. Reporting Adverse Events to the Responsible IEC/IRB and Health Authorities

Adverse events that meet the IEC/IRB requirements for reporting must be reported within the IEC/IRB's written guidelines. Each clinical site will refer to and follow any guidelines set forth by their Approving IEC/IRB. Each clinical site will refer to and follow any guidelines set forth by their local governing Health Authorities.

The Sponsor will report applicable Adverse Events to the local health authorities according the written guidelines, including reporting timelines.

## 13.4.3. Event of Special Interest

None.

## 13.5. Reporting of Pregnancy

Subjects reporting pregnancy (by self-report) during the study will be discontinued after the event is recorded as an Adverse Event. Once discontinued, pregnant participants and their fetuses will not be monitored for study related purposes. At the Investigator's discretion, the study participant may be followed by the Investigator through delivery. However, this data will not be collected as part of the clinical study database. Pregnant participants are not discontinued from contact lens or solution related studies for safety concerns, but due to general concerns relating to pregnancy and contact lens use. Specifically, pregnant women are discontinued due to fluctuations in refractive error and/or visual acuity that occur secondary to systemic hormonal changes, and not due to unforeseen health risks to the mother or fetus.

#### 14. STATISTICAL METHODS

## 14.1. General Considerations

Statistical Analysis will be undertaken by the sponsor or under the authority of the sponsor. A general description of the statistical methods to be implemented in this clinical trial is outlined below. More details will be included in the stand-alone Statistical Analysis Plan (SAP). The SAP will be developed and finalized prior to database lock.

All data summaries and statistical analyses will be performed using the SAS software Version 9.4 or higher (SAS Institute, Cary, NC). Throughout the analysis of data, the results for each subject/eye will be used when available for summarization and statistical analysis. Unscheduled visits will be summarized separately and will be excluded from the statistical analysis.

Summary tables (descriptive statistics and/or frequency tables) will be provided for all baseline variables, efficacy variables and safety variables as appropriate. Continuous variables will be summarized with descriptive statistics (n, mean, standard deviation [SD], median, minimum and maximum). Frequency count and percentage of subjects or eyes within each category will be provided for categorical data.

## 14.2. Sample Size Justification

This study was designed and powered to show non-inferiority of the Test lens compared to the Control lens with respect to logMAR Visual Acuity, Slit Lamp Findings (Grade 3 or higher) and CLUE comfort. It was assumed there was no difference between the Test and Control lens with respect to slit lamp findings and a 1 letter difference (0.02) between the Test and Control lenses with respect to visual acuity logMAR. Based on data from 3 historical studies, it was assumed there was a 2-point difference between the Test and Control lenses with respect to CLUE comfort based on the summary statistics from the first period of the historical studies.

In addition to the endpoints mentioned above, this study was also powered to demonstrate non-inferiority of the Test lens relative to the Control lens with respect to vision satisfaction in bright lighting and the proportion of eyes with acceptable fitting while the Test lens is significantly superior to 90%.

Unless otherwise specified, the sample size was calculated to achieve a statistical power of at least 80% and a type I error of 5%.

A total of 5 historical studies were utilized in the sample size calculation. Table 6 displays the studies, their corresponding study design and the number of subjects enrolled and completed perprotocol.

Table 6: Historical Studies Included in Sample Size Calculation

| Study | Study Design | Endpoints Collected | No.<br>Enrolled | No. Completed<br>Per-Protocol |
|---|---|---|---|---|
| , | | . j | | |
| | 2X3 Crossover | CLUE, SLF Lens Fit | 135 | 132 |
| | 2X3 Crossover | CLUE, Visual Acuity (logMAR), SLF, Lens Fit | 133 | 121 |
| | 2X3 Crossover | CLUE, SLF Lens Fit | 92 | 78 |
| | Single-Arm | SLF, Lens Fit | 54 | 48 |
| | Single-Arm | SLF, Lens Fit | 56 | 41 |

Table 7: Descriptive Summary of CLUE Scores by Domain Pooled Across Historical Studies

| Overall Quality of Vision | 64.49 (17.221) | 64.44 (23.351) |
|---------------------------|----------------|----------------|

<sup>1</sup>SD = Standard Deviation

Table 8: Descriptive Summary of Visual Acuity (logMAR) - 2-Week Follow-up Evaluation-Period 1 only

| Visual Acuity High<br>Illumination High Contrast | Test | Control |
|---|---|---|
| [Mean(SD) <sup>1</sup> ] | -0.088 (0.0.0862) | -0.0622 (0.0740) |

<sup>&</sup>lt;sup>1</sup>SD = Standard Deviation

Table 9: Descriptive Summary of Mechanical Lens Fitting Pooled Across all Historical Studies

| Any Unacceptable Lens Fit <sup>1</sup> [n(%)] | Test n (%) | Control n (%) |
|-----------------------------------------------|------------|---------------|
| Fitting Evaluation | 0(0.0) | 0 (0.0) |
| 2-Week Follow-up | 0 (0.0) | 0 (0.0) |

<sup>&</sup>lt;sup>1</sup>The percent of any unacceptable fit is calculated using Total Unique eyes as a denominator

Table 10: Descriptive Summary of Slit Lamp Findings Pooled Across all Historical Studies

| SLF Grade 2 | Test n (%) | Control n (%) |
|------------------------------|-------------|---------------|
| Corneal Edema | 0 (0.0) | 0 (0.0) |
| Conjunctival Injection | 59 (6.86) | 59 (21.85) |
| Tarsal Abnormalities | 51 (5.93) | 24 (8.89) |
| Corneal Neovascularization | 3 (0.35) | 0 (0.0) |
| Corneal Staining | 3 (0.35) | 0 (0.0) |
| Other Findings | 0 (0.0) | 0 (0.0) |
| Total Eyes (N) | 860 | 270 |
| Any SLF Grade 2 <sup>2</sup> | 116 (13.48) | 83 (33.74) |
| Any SLF Grade 3+ | 0 (0.0) | 0 (0.0) |
| Total Unique Eyes | 860 | 270 |
| Total Unique Subjects | 430 | 135 |

<sup>%=</sup> nx100/N; SD=Standard Deviation

JJVCI CONFIDENTIAL CR-6305, v4.0 Amendment 3.0 

<sup>&</sup>lt;sup>1</sup>All SLF reported for this study are combined for the purposes of summarizing

<sup>&</sup>lt;sup>2</sup> The percent (%) of Any Grade 2 is calculated using the Total Unique Eyes as the denominator

| Questionnaire Item/ Response | Test | Control |
|--------------------------------------------|-------------|-------------|
| Vision Satisfaction in Bright Light [n(%)] | | |
| Strongly Agree | 72 (29.75) | 51 (21.07) |
| Agree | 129 (53.31) | 130 (53.72) |
| Neither Agree Nor Disagree | 24 (9.92) | 21 (8.68) |
| Disagree | 17 (7.02) | 33 (13.64) |
| Strongly Disagree | 0 (0.0) | 7 (2.89) |

#### **CLUE Comfort Scores**

With respect to CLUE comfort, based on historical data from Period 1, a mean difference of 2 points was assumed and a standard deviation of 21, an additive equivalence test in PROC Power for two sample means was used to Test for non-inferiority. A non-inferiority margin of -5 points was used since this is considered to be no more than a 10% shift in the distribution of CLUE scores.

## **Mechanical Lens Fit (Test Lens)**

The estimated sample size to test the primary hypothesis (H0 PT  $\leq$  P0, H1: PT > P0) is 100. The sample size was calculated using PROC POWER for one sample proportion using an exact Test of a Binomial Proportion.

#### Visual Performance (logMAR)

Sample size calculation for visual performance (logMAR) was carried out using an approximation of the power of an F-test derived from the non-centrality parameter calculated form the observed F statistic of a linear model.<sup>8</sup>

#### Model details:

visual performance was analyzed using a linear mixed model. Lens type was included as the only fixed effect. A compound symmetric (CS) covariance matrix was used to model the correlation between measurements on the same subject across study periods. Below is the variance-covariance matrix used in the visual performance model.

$$\sum_{\textit{Visual Acuity}} \begin{pmatrix} 0.004047 & 0.002894 \\ 0.002894 & 0.004737 \end{pmatrix}$$

# **Slit Lamp Findings**

There were no Grade 3 or higher SLFs observed in any of the historical studies. Assuming no difference between study lenses and a correlation 0.70 between left and right eyes within the same subject (intra-subject correlation), a reference rate of no more than 5% was assumed (worse-case scenario) with a non-inferiority odds ratio margin of 2. A total of 2000 replicating trials were simulated, each replicated sample was analyzed using a generalized estimating equation (GEE)

model with a binary distribution and the logit as the link function. Each model included lens type as the only fixed, eye was included as a random effect. The Odds ratio and corresponding 95% confidence interval was used estimate differences between the Test and Control lenses. The upper limit of each 95% confidence interval was compared to 2; if the upper limit was below 2 then NI=1; otherwise NI=0. Statistical power was calculated as the average NI. A sample size of 224 (112 per arm) was chosen to achieve a minimum statistical power of 80%.

Using a reference rate for the control of 5% and no more than a 5% difference between the Test and Control lenses translate to an odds ratio margin of 2. A reference rate of 5% was used as the worst-case scenario.

#### **Individual Questionnaire Items**

Vision satisfaction in bright lighting sample size estimates were calculated using historical data from CR-5960.<sup>7</sup> One-thousand boot strap samples were simulated based on the historical data. For each replicated sample a generalized linear mixed model was used with a multinomial distribution and the cumulative logit as the link function. Lens type was included in the model as the only fixed effect.

Using a reference rate of 50% for the Control lens and assuming no difference between the Test and Control a 10% difference translate to a cumulative odds ratio margin of 0.67. the reference rate of 0.50 was used as the worst-case scenario.

Table 12: Sample Size Estimates and Power Calculations for Primary Endpoints

| Endpoint | Number per<br>Subjects to<br>Complete | Power |
|---|---|---|
| Distance Monocular Visual Acuity (logMAR) | 30 | 86% |
| SLFs (Grade 3 or Higher) | 224 | 80% |
| Acceptable lens Fit (Test Lens Only) | 100 | 82% |
| CLUE Comfort | 224 | 87% |
| Vision Satisfaction in Bright Lighting | 40 | 87% |

Table 13: Sample Size Estimates and Power Calculations for Secondary Endpoints

| Endpoint | Number per Subjects to<br>Complete | Power |
|--------------------------------|------------------------------------|-------|
| CLUE Handling | 224 | 63% |
| CLUE Overall Quality of Vision | 224 | 71% |

As indicated in Table 12 and 13 above, the sample size chosen for this study was primary driven by slit lamp findings (Grade 3 or higher) and overall comfort. The plan is to enroll 236 eligible subjects (118 subject per arm) with a target of 112 subjects to complete each arm in the study. During the enrollment period, the subject drop-out rate with be closely monitored, if an unexpectedly high dropout rate is observed, then the targeted total enrollment number maybe be increased accordingly to ensure that a minimum of 224 subjects complete the study.

## 14.3. Analysis Populations

# **Safety Population:**

All subjects who were administered any test article excluding subjects who drop out prior to administering any test article. At least one observation should be recorded.

## **Per-Protocol Population:**

All subjects who have successfully completed all visits and did not substantially deviate from the protocol as determined by the trial cohort review committee prior to database hard lock (Per-Protocol Population). Justification of excluding subjects with protocol deviations in the per-protocol population set will be documented in a memo to file.

## **Intent-to-Treat (ITT) Population:**

All randomized subjects regardless of actual treatment and subsequent withdrawal from study or deviation from protocol. At least one observation should be recorded.

Safety variables will be summarized on both safety and PP populations whereas efficacy variables will be summarized on the per-protocol and Intent-to-Treat population.

# 14.4. Level of Statistical Significance

All planned analysis for this study will be conducted with an overall type I error rate of 5%.

# 14.5. Primary Analysis

## Primary efficacy analysis:

All the efficacy analyses will be conducted on PP population. As sensitivity analysis, the efficacy analysis will be repeated on the ITT population regardless of missing data.

#### **Visual Acuity**

Distance monocular visual acuity (logMAR) will be tested under bright illumination low contrast conditions at the 2-week follow-up evaluation and will be analyzed using a Bayesian normal random-effects model to compare the Test and Control lenses. The regression model will include lens type as the only fixed effect. Clinical site and subject will be included as random effects. Other subject characteristics such as gender and age will be included as fixed effects when appropriate.

#### The Model:

Let  $y_{ijkl}$  the visual acuity (logMAR) for the  $l^{th}$  subject at the  $k^{th}$  site, assigned to the  $i^{th}$  lens for the  $j^{th}$  eye. The likelihood for  $y_{ijkl}$  is constructed as follows:

$$y_{ijkl} \sim N(\mu_{ijkl}, \sigma_{ijkl}^2)$$

Where,

$$\mu_{ijkl} = \mu_0 + \beta_1 Lens + \gamma_{l(k)} + \alpha_k$$

In this model, lens we define  $Lens_l=0$  for the Control lens and  $Lens_i=1$  for the Test lens. So  $\beta_1$  stands for the difference between the Test and Control lens with respect to logMAR visual performance. A negative  $\beta_1$  indicates the Test performed better than the Control lens.

We assume random subject effects are independent and identically distributed (i.i.d) as  $\gamma_j \sim N(0, \sigma_{subject}^2)$  as random subject and, the random site effect is i.i.d as  $\alpha_k \sim N(0, \sigma_{site}^2)$  for i=1,2 (lens), j=1, 2 (eye), k=1, 2, 3, 4, 5, 6 (site).

For the  $\beta$  coefficients, independent non-informative priors N(0, 1000) will be used. For the variance of random effects  $\sigma_{eye}^2$  and  $\sigma_{site}^2$  independent non-informative conjugate priors inverse-gamma(0.001, 0.001) will be used. For  $\sigma_{ijkl}^2$ , non-informative conjugate priors inverse-gamma(0.001, 0.001) will be used where  $\sigma_{ijkl}^2$ , is the variance of  $y_{ijkl}$ . The metropolis sampler algorithm as implemented in the SAS/STAT MCMC 14.2 procedure will be used to estimate the posterior distribution of the unknown parameters. Inferences will be made based on the 95% posterior credible intervals for relevant parameters.

## **Hypothesis Testing**

The null and alternative hypothesis for visual acuity (logMAR) to test for non-inferiority of the Test lens relative to the Control lens is as follows:

$$H_o: \beta_1 \ge 0.05$$
  
 $H_A: \beta_1 < 0.05$ 

Non-inferiority will be declared if the upper limit of the 95% credible interval of the difference between the Test and Control is below 0.05, i.e.  $P(\beta_1 < 0.05) \ge 0.975$ .

# **CLUE Overall Comfort**

CLUE Comfort scores will be analyzed using a Bayesian normal random-effects model to compare the Test and Control lenses at the 2-week follow-up evaluation. The regression model will include baseline CLUE comfort scores and lens type as fixed effects. Clinical site will be included as random effects. Other subject characteristics such as age, gender, race and iris category will be included as fixed covariates when appropriate.

## The Model:

Let  $y_{ijkl}$  denote the CLUE Comfort score for the  $k^{th}$  subject at the  $j^{th}$  site, assigned to the  $i^{th}$  lens. The likelihood for  $y_{ijkl}$  is constructed as follows:

$$y_{ijkl} \sim N(\mu_{ijkl}, \sigma_{ijkl}^2)$$

Where

$$\mu_{ijkl} = \mu_0 + \beta_1 Lens + \beta_2 baseline + \gamma_k$$

In this model, we define Lens=0 for the Control lens and Lens = 1 for the Test lens. So  $\beta_1$  stands for the difference between the Test and Control lens with respect to CLUE comfort; A positive  $\beta_1$  indicates the Test performed better than the Control.

We assume random site effects are independent and identically distributed (i.i.d) as  $\gamma_j \sim N(0, \sigma_{site}^2)$  for site for i=1, 2 (lens), j=1, 2, 3, 4, 5, 6 (site), k=1....n (subject/site).

For the  $\beta$  coefficients, independent non-informative priors N(0, 1000) will be used. For the variance of random effect of  $\sigma_{site}^2$  an independent non-informative conjugate prior, inverse-gamma

(0.001, 0.001) will be used. Starting values for the mean and variance of CLUE scores will be 60 and 400 (since standard deviation of CLUE is normalized to be 20), respectively. The Metropolis sampler algorithm as implemented in the SAS/STAT MCMC 14.2<sup>14</sup> procedure will be used to estimate the posterior distribution of the unknown parameters. Inferences will be made based on the 95% posterior credible intervals for relevant parameters.

# Hypothesis Testing

The null and alternative hypotheses for CLUE comfort non-inferiority of the Test lens relative to the Control lens are as follows:

$$H_o$$
:  $\beta_1 \leq -5$ 

$$H_A: \beta_1 > -5$$

Non-inferiority will be declared if the lower bound of the 2-sided 95% credible interval of the difference between the Test lens and the Control lens is greater than -5, i.e.,  $P(\beta_1 > -5) \ge 0.975$ .

# **Vision Satisfaction in Bright Lighting**

Vision satisfaction in bright lighting at the 2-week follow-up evaluation will be analyzed using a Bayesian multinomial model for ordinal data. The regression model will include lens type as the only fixed effect. Clinical site will be included as a random effect. Other subject characteristics such as age, gender, race and iris category will be included when appropriate.

#### The Model:

Let  $y_{ijk} = (y_{ijk1}, y_{ijk2}, y_{ijk3}, y_{ijk4}, y_{ijk5})$  denote the rating for the  $k^{th}$  subject, from the  $j^{th}$  site, assigned to the  $i^{th}$  study lens. Possible values of  $y_{ijk}$  are 1 if the subject rating of vision satisfaction in bright lighting are X and 0 otherwise (x=1 for Strongly Agree and X=5 for Strongly Disagree, respectively). The likelihood is constructed as follows:

$$\begin{aligned} y_{ijk} \sim & \text{Multinomial } (P_{ijk1}, \ P_{ijk2} \ , P_{ijk3}, P_{ijk4}, P_{ijk5}) \\ P_{ijk1} &= \gamma_{ijk1} \\ P_{ijkX} &= \gamma_{ijkX} - \gamma_{ijk(X-1)} \ 2 \leq n \leq 4 \\ P_{ijk5} &= 1 - \sum_{x=1,...4} P_{ijkX} \end{aligned}$$

$$Logit(\gamma_{ijklmX}) = \theta_n + \beta_1 Lens + \gamma_j$$

Where  $\theta_n$  is the intercept for levels n=1,2,3,4,  $P_{ijk1} = \Pr(\gamma_{ijk1} = 1)$  with respect to the vision satisfaction in bright lighting item. We assume the random clinical site effects are i.i.d as  $\gamma_j \sim N(0, \sigma_{site}^2)$  for i=1,2 (lens), j=1, 2, 3, 4, 5, 6(site) and k=1,....n (subject/site)

In this model, the lens I will be determined by the period j and sequence k, therefore i is denoted as a function of j and k. We define  $Lens_i=0$  for the Control lens and  $Lens_i=1$  for the Test lens.

Independent vague N(0, 1000) priors for the regression coefficients  $\beta_i$  i=1,...5. For  $\theta_n$ , we are considering the following priors

$$\begin{split} &\pi 0(\theta 1) \sim N(0,\!100) \\ &\pi 0(\theta 2|\, \theta 1) \sim N(0,\!100) I(\theta \!\!>\!\! \theta 1) \\ &\pi 0(\theta 3|\, \theta 2) \sim N(0,\!100) I(\theta \!\!>\!\! \theta 2) \\ &\pi 0(\theta 4|\, \theta 3) \sim N(0,\!100) I(\theta \!\!>\!\! \theta 3) \end{split}$$

For the variance of random effects independent vague normal priors will also be used;  $\sigma_s^2$  ~inverse-gamma(0.001, 0.001). The Metropolis sample algorithm as implemented in the SAS/Stat MCMC Procedure will be used to estimate the posterior distributions of the unknown parameters. Inferences will be made based on the posterior credible interval for the relevant parameters.

# **Hypothesis Testing**

The null and alternative hypotheses for non-inferiority are as follows:

$$H_o: p_t - p_c \le -0.1$$
  
 $H_A: p_t - p_c \ge -0.1$ 

where  $p_T$  and  $p_C$  are the proportions of patients with positive response (agree or strongly agree) in Test group and Control group, respectively. Non-inferiority will be established if the lower limit of the 2-sided 95% credible interval of the difference  $(p_T - p_C)$  is above -0.1 (i.e.  $P(p_t - p_c) > 0.1 | data) \ge 0.975$ .

## **Primary Safety Analysis:**

Safety analysis will be conducted on safety population by treatment actually received by subjects.

#### **Acceptable Lens Fit:**

Acceptable lens fit will be analyzed using a Bayesian beta-binomial models for correlated binary data. The regression model will include lens type as the only fixed effects

#### The Model:

Let Y1 and Y2 denote the binary outcomes of acceptable lens fit for the left and right eyes, respectively, when wearing the test lens. Considering the correlation,  $\rho$ , between Y1 and Y2, the distribution of the sum Y = Y1 + Y2 is obtained by the mixture of two variables. One of them follow a binomial distribution Bin(2, p) with mixing probability (1-p) and the other one follows a modified Bernoulli distribution MBern(p), taking value 0 and 2 rather than conventional 0 and 1, with mixing probability p:

$$P(Y=y|\ p,\ \rho)=(1-\rho)Bin(2,\ p)I_{A1}+\ \rho MBern(p)I_{A2}$$
 Where  $I_{A1}=\{0,\ 1,\ 2\}$  and  $I_{A2}=\{0,\ 2\}$ 

To overcome the complexity of the mixture likelihood a latent variable  $Z_i$ , i = 1, 2 is introduced in the model to indicate in which component of the model the observation  $y_i$ , i=1, 2, belongs to, that is,

$$z_i = \begin{cases} 1, & \text{if the observation belong to the MBern(p),} \\ 0, & \text{if the observation belong to the Bin(2, p)} \end{cases}$$

The joint distribution of the augmented data (Yi, Zi), i=1, 2, is given by

$$P(Y=y_i,Z=z_i|\;p,\rho)=\;\;\rho^{z_i}p^{y_iz_i/2}(1-p)^{(2-y_i)z_i/2}(1-\rho)^{1-z_i}\binom{2}{y_i}p^{y_i(1-z_i)}(1-p)^{(2-y_i)(1-z_i)}$$

The posterior distribution of  $(p, \rho)$  given (y, z) is

$$P(p, \rho | \mathbf{z}, \mathbf{y}) = P(\mathbf{y}, \mathbf{z} | p, \rho) \pi_0(p, \rho),$$

Where,  $\pi_0$  is joint prior distribution of  $(p, \rho)$ . Here we assume p and  $\rho$  to be independent with a prior beta $(\alpha,\beta)$  for p and uniform(0,1) for  $\rho$ . Hence the joint distribution of  $(p, \rho)$  is given by  $\pi_0(p, \rho) \propto p^{\alpha-1}(1-p)^{\beta-1}$ . The Metropolis sampler algorithm as implemented in the SAS/STAT MCMC Procedure will be used to estimate the posterior distributions of the parameters  $(p, \rho)$ . Inferences will be made based on a posterior credible interval for the relevant parameters.

# **Hypothesis Testing**

With respect to Acceptable lens fit the null and alternative hypothesis for superiority is as follows:

$$H_0 = p_T \le 0.90$$
  
 $H_1 = p_T > 0.90$ 

Where,  $p_T$  represents the proportion of subject eyes that achieve acceptable fit for the Test lens. Success for acceptable fit will be declared if the lower bound of the 2-sided 95% credible interval of the proportion is greater than 0.90; i.e.  $P(p_T > 0.90) \ge .975$ .

If the full planned model fails to converge, reduced versions may be considered.

#### **Slit Lamp Findings**

Grade 3 or higher slit lamp findings will be analyzed using a Bayesian Logistic regression randomeffects model to compare the Test and Control lenses. The regression model will include baseline slit lamp findings and lens type. Site and subject will be included in the model as random effects.

Let  $y_{ijkl}=1$  if a Grade 3 or higher SLF is observed and  $y_{ijk}=0$  otherwise for the  $l^{th}$  subject, from the  $k^{th}$  site, assigned to the  $i^{th}$  study lens for the  $j^{th}$  eye.

$$y_{ijkl} \sim Binary(p_{ijkl})$$

$$p_{ijkl} = \frac{\exp(\beta_0 + \beta_1 Lens + \beta_2 Baseline \, SLF_l + \gamma_k + \delta_l)}{1 + \exp(\beta_0 + \beta_1 Lens + \beta_2 Baseline \, SLF_l + \gamma_k + \delta_l)}$$

We assume the random effect for subject are i.i.d as  $\delta_l \sim N(0, \sigma_{subject/site}^2)$  for the random for clinical site are i.i.d as  $\gamma_k \sim N(0, \sigma_{site}^2)$  for i=1,2 (lens), j=1, 2 (eye), k=1, 2, 3, 4, 5, 6 (site) and l=1,...n (subject/site).

In this model, we define  $Lens_i$ =0 for the Control lens and  $Lens_i$ =1 for the Test lens. For the  $\beta$  coefficients, independent non-informative priors N(0, 10000) will be used. For the variance of random effects of  $\sigma_{\text{subject}}^2$  and  $\sigma_{\text{site}}^2$ , independent non-informative conjugate priors inverse-gamma (0.001, 0.001) will be used. The Metropolis-Hastings algorithm as implemented in the SAS/STAT 14.2 PROC MCMC procedure will be used to estimate posterior distributions of the unknown parameters. Inferences will be made based on the posterior credible interval for the relevant parameters.

## **Hypothesis Testing**

The null and alternative hypothesis for Non-inferiority is as follows:

$$\begin{split} H_0 &= p_T - \ p_C \geq 0.05 \\ H_1 &= p_T - \ p_C < 0.05 \ , \end{split}$$

where  $p_T$  and  $p_C$  are the proportions of Grade 3 or higher SLFs in Test group and Control group, respectively.

Non-inferiority will be established if the upper limit of the 2-sided 95% credible interval of the difference  $(p_T - p_C)$  is below 0.05(i.e.  $p(p_T - p_C < 0.05|data) \ge .975$ ).

If the full planned model fails to converge, reduced versions may be considered. In the event that the number of Grade 3 or higher SLFs is too small Grade 2 or higher SLFs will be analyzed and tested as described above.

#### 14.6. Secondary Analysis

**Secondary efficacy analysis:** 

#### **CLUE Overall Quality of Vision and Handling**

CLUE Overall Quality of Vision and Handling will be analyzed using the same statistical method described for CLUE Overall Comfort

#### Secondary safety analysis:

Not Applicable

#### 14.7. Other Exploratory Analyses

Not applicable.

# 14.8. Interim Analysis

There will not be an interim analysis performed on this study.

# 14.9. Procedure for Handling Missing Data and Drop-Outs

Missing or spurious values will not be imputed. The count of missing values will be included in the summary tables and listings.

Subject dropout is expected to be one of the main reasons of missing data in this clinical trial. Past clinical trials don't provide the evidence that subject dropout is systematic or not-at-random. To evaluate the impact of missing data, sensitivity analysis may be considered by automatically sampling all missing values and incorporating them in the Markov chain for the parameters using the PROC MCMC procedure.

# 14.10. Procedure for Reporting Deviations from Statistical Plan

The analysis will be conducted according to that specified in above sections. There are no known reasons for which it is planned to deviate from these analysis methods. If for any reason a change is made, the change will be documented in the study report along with a justification for the change.

#### 15. DATA HANDLING AND RECORD KEEPING/ARCHIVING

# 15.1. Electronic Case Report Form/Data Collection

The data for this study will be captured on electronic case report forms (eCRFs) using an EDC system (BioClinica). An authorized data originator will enter study data into the eCRFs using the EDC system. Data collected on equipment that is not captured in EDC will be formatted to the specification of the JJVCI database manager and sent to JJVCI for analysis.

External Date Sources for this study include: Not Applicable

The clinical data will be recorded on dedicated eCRFs specifically designed to match the study procedures for each visit. Once completed, the eCRFs will be reviewed for accuracy and completeness and signed by the Investigator. The sponsor or sponsor's representatives will be authorized to gain access to the subject recordation for the purposes of monitoring and auditing the study.

Edit checks, electronic queries, and audit trails are built into the system to ensure accurate and complete data collection. Data will be transmitted from the clinical site to a secure central database as forms are completed or updated, ensuring information accuracy, security, and confidentiality. After the final database lock, the Investigator will be provided with Individual Patient Profiles (IPP) including the full audit trail on electronic media in PDF format for all of the study data. The IPP must be retained in the study files as a certified copy of the source data for the study.

The content and structure of the eCRFs are compliant with ISO14155:2011.<sup>1</sup>

#### 15.2. Subject Record

At a minimum, subject record should be available for the following:

• subject identification

- eligibility
- study identification
- study discussion
- provision of and date of informed consent
- visit dates
- results of safety and efficacy parameters as required by the protocol
- a record of all adverse events
- follow-up of adverse events
- medical history and concomitant medication
- test article receipt/dispensing/return records
- date of study completion
- reason for early discontinuation of test article or withdrawal from the study, if applicable

The subject record is the eCRF or an external record. The author of an entry in the subject record must be identifiable. The first point of entry is considered to be the source record.

Adverse event notes must be reviewed and initialed by the Investigator.

#### 16. DATA MANAGEMENT

#### 16.1. Access to Source Data/Document

The Investigator/Institution will permit trial-related monitoring, audits, IEC/IRB review and regulatory inspection(s) by providing direct access to source data/documents. Should the clinical site be contacted for an audit by an IEC/IRB or regulatory authority, JJVCI must be contacted and notified in writing within 24 hours.

# 16.2. Confidentiality of Information

Information concerning the investigational product and patent application processes, scientific data or other pertinent information is confidential and remains the property of JJVCI. The Investigator may use this information for the purposes of the study only. It is understood by the Investigator that JJVCI will use information developed in this clinical study in connection with the development of the investigational product and therefore may disclose it as required to other clinical investigators and to regulatory agencies. In order to allow the use of the information derived from this clinical study, the Investigator understands that he/she has an obligation to provide complete test results and all data developed during this study to the Sponsor.

#### 16.3. Data Quality Assurance

Steps will be taken to ensure the accuracy and reliability of data, include the selection of qualified investigators and appropriate clinical sites and review of protocol procedures with the Principal Investigator. The Principal Investigator, in turn, must ensure that all Sub-Investigators and clinical site personnel are familiar with the protocol and all study-specific procedures and have appropriate knowledge of the study article.

Training on case report form completion will be provided to clinical site personnel before the start of the study. The Sponsor will review case report forms for accuracy and completeness remotely during the conduct of the study, during monitoring visits, and after transmission to data management. Any data discrepancies will be resolved with the Investigator or designee, as appropriate.

Quality Assurance representatives from JJVCI may visit clinical sites to review data produced during the study and to access compliance with applicable regulations pertaining to the conduct of clinical trials. The clinical sites will provide direct access to study-related source data/documents and reports for the purpose of monitoring and auditing by JJVCI and for inspection by local and regulatory authorities.

#### 17. MONITORING

The study monitors will maintain close contact with the Principal Investigator and the Investigator's designated clinical site personnel. The monitor's responsibilities will include:

- Ensuring that the investigation is being conducted according to the protocol, any subsequent amendments, and regulatory requirements are maintained
- Ensuring the rights and wellbeing of subjects are protected
- Ensuring adequate resources, including facilities, laboratories, equipment, and qualified clinical site personnel
- Ensuring that protocol deviations are documented with corrective action plans, as applicable
- Ensuring that the clinical site has sufficient test article and supplies
- Clarifying questions regarding the study
- Resolving study issues or problems that may arise
- Reviewing of study records and source documentation verification in accordance with the monitoring plan

#### 18. ETHICAL AND REGULATORY ASPECTS

## 18.1. Study-Specific Design Considerations

Potential subjects will be fully informed of the risks and requirements of the study and, during the study, subjects will be given any new information that may affect their decision to continue participation. Subjects will be told that their consent to participate in the study is voluntary and may be withdrawn at any time with no reason given and without penalty or loss of benefits to which they would otherwise be entitled. Only subjects who are fully able to understand the risks, benefits, and potential adverse events of the study, and provide their consent voluntarily will be enrolled.

# 18.2. Investigator Responsibility

The Principal Investigator is responsible for ensuring that the clinical study is performed in accordance with the signed agreement, the investigational plan, Section 4 of the ICH E6 guidelines on Good Clinical Practice (GCP),<sup>2</sup> and applicable regulatory requirements. GCP is an international

ethical and scientific quality standard for designing, conducting, recording, and reporting studies that involve the participation of human subjects. Compliance with this standard provides public assurance that the rights, safety, and well-being of study subjects are protected, consistent with the principles of the Declaration of Helsinki 64<sup>th</sup> WMA General Assembly 2013<sup>3</sup> and that the clinical study data are credible. The Investigator must maintain clinical study files in accordance with Section 8 of the ICH E6 guidelines on Good Clinical Practice (GCP),<sup>2</sup> and applicable regulatory requirements.

## 18.3. Independent Ethics Committee or Institutional Review Board (IEC/IRB)

Before the start of the study, the Investigator (or Sponsor when applicable) will provide the IEC/IRB with current and complete copies of the following documents (where applicable):

- Final protocol and, if applicable, amendments
- Sponsor-approved informed consent form (and any other written materials to be provided to the subjects)
- Investigator's Brochure (or equivalent information) and amendments
- Sponsor-approved subject recruitment materials
- Information on compensation for study-related injuries or payment to subjects for participation in the study
- Investigator's curriculum vitae, clinical licenses, or equivalent information (unless not required, as documented by IEC/IRB)
- Information regarding funding, name of the Sponsor, institutional affiliations, other potential conflicts of interest, and incentives for subjects
- Any other documents that the IEC/IRB requests to fulfill its obligation

This study will be undertaken only after IEC/IRB has given full approval of the final protocol, amendments (if any), the informed consent form, applicable recruiting materials, and subject compensation programs, and the Sponsor has received a copy of this approval. This approval letter must be dated and must clearly identify the documents being approved.

During the study, the Investigator (or Sponsor when applicable) will send the following documents to the IEC/IRB for their review and approval, where appropriate:

- Protocol amendments
- Revision(s) to informed consent form and any other written materials to be provided to subjects
- If applicable, new or revised subject recruitment materials approved by the Sponsor
- Revisions to compensation for study-related injuries or payment to subjects for participation in the study
- Investigator's Brochure amendments or new edition(s)
- Summaries of the status of the study (at least annually or at intervals stipulated in guidelines of the IEC/IRB)
- Reports of adverse events that are serious, unanticipated, and associated with the test articles, according to the IRB's requirements
- New information that may adversely affect the safety of the subjects or the conduct of the study
- Major protocol deviations as required by the IEC/IRB

- Report of deaths of subjects under the Investigator's care
- Notification if a new Investigator is responsible for the study at the clinical site
- Any other requirements of the IEC/IRB

For protocol amendments that increase subject risk, the amendment and applicable informed consent form revisions must be submitted promptly to the IEC/IRB for review and approval before implementation of the change(s).

At least once a year, the IEC/IRB will review and reapprove this clinical study. This request should be documented in writing.

At the end of the study, the Investigator (or Sponsor where required) will notify the IEC/IRB about the study completion. Documentation of this notification must be retained at the clinical site and a copy provided to the CRO or Sponsor as applicable.

#### 18.4. Informed Consent

Each subject must give written consent according to local requirements after the nature of the study has been fully explained. The consent form must be signed before performance of any study-related activity. The consent form that is used must be approved by both the Sponsor and by the reviewing IEC/IRB. The informed consent is in accordance with principles that originated in the Declaration of Helsinki,<sup>3</sup> current ICH<sup>2</sup> and ISO 14155<sup>1</sup> guidelines, applicable regulatory requirements, and Sponsor Policy.

Before entry into the study, the Investigator or an authorized member of the clinical site personnel must explain to potential subject the aims, methods, reasonably anticipated benefits, and potential hazards of the study, and any discomfort it may entail. Subjects will be informed that their participation is voluntary and that they may withdraw consent to participate at any time.

The subject will be given sufficient time to read the informed consent form and the opportunity to ask questions. After this explanation and before entry into the study, consent should be appropriately recorded by means of the subject's dated signature. After having obtained the consent, a copy of the informed consent form must be given to the subject.

# 18.5. Privacy of Personal Data

The collection, processing and disclosure of personal data and medical information related to the Study Subject, and personal data related to Principal Investigator and any clinical site personnel (e.g., name, clinic address and phone number, curriculum vitae) is subject to compliance with the Health Information Portability and Accountability Act (HIPAA) in the United States<sup>11</sup> and other applicable personal data protection and security laws and regulations. Appropriate measures will be employed to safeguard these data, to maintain the confidentiality of the person's related health and medical information, to properly inform the concerned persons about the collection and processing of their personal data, to grant them reasonable access to their personal data and to prevent access by unauthorized persons.

All information obtained during the course of the investigation will be regarded as confidential. All personal data gathered in this trial will be treated in strictest confidence by Investigators,

monitors, Sponsor's personnel and IEC/IRB. No data will be disclosed to any third party without the express permission of the subject concerned, with the exception of Sponsor personnel (monitor, auditor), IEC/IRB and regulatory organizations in the context of their investigation related activities that, as part of the investigation will have access to the CRFs and subject records.

The collection and processing of personal data from subjects enrolled in this study will be limited to those data that are necessary to investigate the efficacy, safety, quality, and utility of the investigational product(s) used in this study.

These data must be collected and processed with adequate precautions to ensure confidentiality and compliance with applicable data privacy protection laws and regulations.

The Sponsor ensures that the personal data will be:

- processed fairly and lawfully
- collected for specified, explicit, and legitimate purposes and not further processed in a way incompatible with these purposes
- adequate, relevant, and not excessive in relation to said purposes
- accurate and, where necessary, kept current

Explicit consent for the processing of personal data will be obtained from the participating subject before collection of data. Such consent should also address the transfer of the data to other entities and to other countries.

The subject has the right to request through the Investigator access to his personal data and the right to request rectification of any data that are not correct or complete. Reasonable steps should be taken to respond to such a request, taking into consideration the nature of the request, the conditions of the study, and the applicable laws and regulations.

Appropriate technical and organizational measures to protect the personal data against unauthorized disclosures or access, accidental or unlawful destruction, or accidental loss or alteration must be put in place. Sponsor personnel whose responsibilities require access to personal data agree to keep the identity of study subjects confidential.

#### 19. STUDY RECORD RETENTION

In compliance with the ICH/GCP guidelines,<sup>2</sup> the Investigator/Institution will maintain all CRFs and all subject records that support the data collected from each subject, as well as all study documents as specified in ICH/GCP<sup>2</sup> and all study documents as specified by the applicable regulatory requirement(s). The Investigator/Institution will take measures to prevent accidental or premature destruction of these documents.

Essential documents must be retained until at least two (2) years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region or until at least two (2) years have elapsed since the formal discontinuation of clinical development of the investigational product. These documents will be retained for a longer period if required by the applicable regulatory requirements or instructed by

the Sponsor. It is the responsibility of the Sponsor to inform the Investigator/Institution as to when these documents no longer need to be retained.

If the responsible Investigator retires, relocates, or for other reasons withdraws from the responsibility of keeping the study records, custody must be transferred to a person who will accept the responsibility. The Sponsor must be notified in writing of the name and address of the new custodian. Under no circumstance shall the Investigator relocate or dispose of any study documents before having obtained written approval from the Sponsor.

If it becomes necessary for the Sponsor or the appropriate regulatory authority to review any documentation relating to this study, the Investigator must permit access to such reports. If the Investigator has a question regarding retention of study records, he/she should contact JJVCI.

#### 20. FINANCIAL CONSIDERATIONS

Remuneration for study services and expenses will be set forth in detail in the Clinical Research Agreement. The Research Agreement will be signed by the Principal Investigator and a JJVCI management representative prior to study initiation.

JJVCI reserves the right to withhold remuneration for costs associated with protocol violations such as:

- Continuing an ineligible subject in the study
- Scheduling a study visit outside the subject's acceptable visit range

JJVCI reserves the right to withhold final remuneration until all study related activities have been completed, such as:

- Query resolution
- Case Report Form signature
- Completion of any follow-up action items

#### 21. PUBLICATION

This study will be registered on ClinicalTrials.gov by the Sponsor.

#### 22. REFERENCES

- 1. ISO 14155:2011: Clinical investigation of medical devices for human subjects Good clinical practice.
- 2. International Conference on Harmonization Good Clinical Practice E6 (ICH-GCP): <a href="http://www.ich.org/products/guidelines/efficacy/article/efficacy-guidelines.html">http://www.ich.org/products/guidelines/efficacy/article/efficacy-guidelines.html</a>
- 3. Declaration of Helsinki Ethical principles for Medical Research Involving Human Subjects. <a href="http://www.wma.net/en/30publications/10policies/b3/index.html">http://www.wma.net/en/30publications/10policies/b3/index.html</a>.
- 4. United States (US) Code of Federal Regulations (CFR). In <a href="https://www.gpo.gov/fdsys/browse/collectionCfr.action?collectionCode=CFR">https://www.gpo.gov/fdsys/browse/collectionCfr.action?collectionCode=CFR</a> (Ed.).

| 5. | Buch, J. |
|-----|-----------------------------------------------------------------------|
| | Design Validation of senofilcon A with New UV-blocking Additive. 2018 |
| 6. | Buch, J. O. Clinical Evaluation of Test |
| | Lenses Manufactured with Different Curing Methods. 2017 |
| 7. | Buch, J. Evaluation of Approved |
| | and Investigational Contact Lenses. 2018 |
| 8. | Buch, J. Contact Lenses with New |
| | UV-blocker Manufactured with Different Techniques. August 01, 2018 |
| 9. | Buch, J. Diagnostic Contact Lens |
| | Fitting with new UV-blocker Prototype: Study 1.April 24 2018 |
| 10. | Buch, J. Diagnostic Contact Lens |
| | Fitting with new UV-blocker Prototype: Study 2.May 08 2018 |
| 11. | Health Information Portability and Accountability Act (HIPAA). In |
| | https://www.hhs.gov/hipaa/for-professionals/privacy/index.html (Ed.). |

| APPENDIX A: PATIENT REPORTED OUTCOMES (STUDY QUESTIONNAIRES) |
|--------------------------------------------------------------|

| Protocol 6305 | Johnson & Johnson Vision Care, Inc. | Confidential |
|---------------|-------------------------------------|--------------|

| Protocol 6305 | Johnson & Johnson Vision Care, Inc. | Confidential |
|---------------|-------------------------------------|--------------|

| ADDENIDIY I | D. DATIENT | INSTRUCTION | CHIDE |
|-------------|------------|-------------|---------|
| APPENDIX | B: PAIIKNI | INSTRUCTION | CTUII)K |

A Patient Instruction Guide will be provided separately.
# APPENDIX C: PACKAGE INSERT (APPROVED PRODUCT) ACUVUE OASYS®

I vision is acceptable, perform a silt tamp examination to assess adequate il premision and involvente. Il it is a compatible, disposas the involve industrial the patient to refusit is now veek for massessment (see disposaing and following information in PATENT MAMAGRART).

All potents should be suggled with a copy of the PATRAT BASTRUCTION OLDE for these feness. Copies are available for download at wave.acutes.com.

# TORIC FITTING GUIDELINES

Although most season of the filter procedure are the rigid for all post of an all the control of the filter procedure are the rigid for the post of the filter and the control of the filter and the proper of at their dense, and the filter an instance for the proper of at their dense, and the filter procedure of the filter and their procedure dense are the stable, and the filter dense are the system of dense are the stable and the filter dense and the system of the filter and the filter dense are the system of the filter and the filter dense dense and the system of the filter and the fi

In termine the description of the total term, you'll be the proposed of the state o

where where we have the color 200 beauties the count promotion in particular the color 200 beautiful to 200 beautiful to 200

After the patient's parkmease under the above conditions in contributed teams of student stocks or parkmease, the above conditions or incoherancy distributes a stock parkmease, and a parkmease and a parkmea

Manifest described galaction alread for another sinds entirely pre-mained entered galaction alread for another sinds and another sinds and the Admirition of the greatest on terms and alread sinds of an experiment of the sinds of these specimens may lake a possible of the sinds of the sinds of the sinds of these specimens may lake a possible shade on the transmission of the sinds of these specimens may be a possible of the sind of the structural and advantage. The sinds of the sinds of the sinds of the transmission of the sinds of t

The many our publics consider that only applicable to the control of the control our control of the control our control of the control our control of the control our control of the control our control our control of the control our control of the control our

The studies is lessed to the persons of the persons of the studies is lessed to the persons of the studies. The studies is sent the studies of the studies o

One of the part of

New York of the Commission on the Hospital Could in America (1986) with a concentration on a first source (1986) with a concentration on a first source (1986) with a concentration of the concentrati

REPLACEMENT SCHEDULE

(1) This has beque to additional following that recommendate for

(1) Challed and the third process of the control of the cont


A figure of the rest power of the level board or the patient's ACO may are
ACO. 2010; s. 1.5 are set "Office and Office are now here
3. About the area is entire for a minimum for the rest in the area of t

LENS CARE DIRECTIONS
There are decread to a Tar Care Primitive doubt problem promote deviation of the Care Primitive doubt problem promote deviation of the Care Primitive deviation of the Care Primitive deviation of the respect of the deviation of the respect of the care promoted problem. The Care Primitive deviation of the Care Primitive deviation

The complete retention concentry or other two two-flowing data-for complete retention concentry or other two two-flowing data-ing metables for channels are accounted. The forest retention of the concentration of the c

HOW SUPPLIED

Each sense hour is expected as Leaved Leaven Expect contemp belomed among such as the residence of the sense of the contemp contemp belomed with such such contemp leaven and the sense of

REPORTING OF ADVERSE REACTIONS



Althouse & Johnson & Johnson Ware Care Companies 2015.

By Where & Johnson Waier Care Gallerine & Advance Water Care Person & Land March Care Person & Advance Water Care Person & Person March 11 (2017). Advance March 11 (2017).

Faultion marcher Although Care Person & Person Care Care Person Per

ACLAUE DASTIF and HTDRACLEAP are troberrats of Johnson & Johnson Wein Cass Companies.

# MONOVISION FITTING GUIDELINES

Mexical 2, Contrain which you all congress designment with human Auditors in since Albert and another selection with the excession and COA in the COA one you off their design consistent with the COA one you off their design Coamment (COA one you off their design of the COA one you off their design Coamment and their design of their design of their design of their method selection and their design of their design of Orac method selection and one of their design of Orac method selection and one of their design of Orac method selection and one of the coamment of Orac method selection and one of the coamment of Orac method selection and one of Orac method selection and one of Orac method selection and one of Orac method selection and Orac method selection

1. visually demanding abundons such on operating intensibly designation metabour a profession and the control benefits and control of the con

O Wante Demondration of the properties of the pr A distance of a reasonable season to consist a figure of the control of the contr

When ADD research control is the second of t

iMPORTME. Please read carefully and keep this immunifies for kindmunifier for kindmunifier and kindmunifier the kindmunifier are kind glode is interred for the type. Care Professional, but should be made available to patient any open request.

The Syn Care Professional should provide the patients with the appropriate for successional should provide the patients with the appropriate for successional should provide the patients with the appropriate for the professional should provide the patients of any properties for the professional states.

ACUVULE CONTROLL LENS ES ACUVIE COARTS BEAND CONTROLL LENS ES ACUVIE COARTS BEAND CONTEXT LENS ES ACUVIE COARTS BEAND CONTEXT LENS FOR ACUVIE COARTS BEAND CONTEXT LENS FOR ACUVIE COARTS FROM CONTEXT LENS FOR PERSENCEDA

serofficon A Sort (hydrophilic) Contact Lensel Visibility Thried with UV Blocker for Dally and Extended Wear

ROW Sale Dry or on the order of a Romand practicion

# SYMBOLS KEY

The following symbols may appear on the label or certain.

| ET MISIOL | ABOL DEFINITION |
|---|---|
| All | Consult Instructions for Use |
| 1 | Manufactured by or in |
| บ | Date of Manufacture |
| 04 | Use By Date (repression date) |
| COL | Batch Code |
| Ī | Sterile Using Sharm or Dry Heat |
| ERA | Dismetor |
| 36 | Babe Curve |
| 0 | Diopter (lens power) |
| F) | Ophodie |
| ARS | Auto |
| MAX ADD | Near ADD |
| tow | "Low" Near ADD |
| OW | "Mediun" New ADD |
| HEH | "High" Neer ADD |
| 100 | Quality System Cartification Symbol |
| - Land | UN-Blocking |
| 0 | Fee Paid for Waste Management |
| <b>8</b> ,00 | CAUTICINE U.S. Federal law restricts this device to sale by or on the order of a loomed practitions: |
| 0 | Lana Chartadon Cornet |

Crientation Procreet (Lens Inside Out)

Date on Multi-Purpose Solution Bottle

Librard any invarient problem after the reconstruction between the table of court and a problem of the court table of court flames, courted flames, the problem of the prob

We recovered to the control of the c

Lear Permission of creativities are here for it is a few LMB angue of 500 mmb.

Lear Permission and the second control of the erons are traind than using Possible (Baie Dye 84 to make the forone more intending. A becausings) at Underdring monomer is used to those U.

m has the control of



on data san statural bar mandament isken frough the cartral 3,4 mil parties for the first and state of the cartral 3,5 mil parties for the first and state of the cartral 3,5 mil parties for

The second of the second of th

numberoe d'une derition an less tray 1% in the UNB rarge of 200 ran to and less than 10% in the UNA rarge of 316 ran to 300 ran for the entire

NOTE Lang-latra exposure to VV radiation is one of the risk lisetars associated with classifier. In case, the second control of control of process is based on marrier of stori on such as revenements confidence identice, geography, storic cover language parassociate in the storic as a fundamental professional procession against humal by Viraliania, Viraliania, viraliania, the second procession against humal by viraliania.

specificially indicated on product lickeling for sum in both host and democal

Anny and earth very explore come audions on the common terms

Do not drow in addition after a considerable in the first sum of contact lines

Anny as the common after a contact lines and the first sum of contact lines

Anny as the contact in the positions trent for the sum of contact lines

and form.

To see the democratic sum of the contact such as the contact contact lines

To see the democratic sum of the contact such as the contact contact lines

To see the democratic sum of the contact such that the contact contact lines

To see the contact contact such as the contact model and the see

To see the contact contact such as the contact model and see the

To contact on an or exploration and the time terms are contact to the contact model as seen and and one of the contact contact in the contract model as seen and the contact and the contact contact in the contract contact and are as a section of the contact contact and are as a section of the contact contact and are as a section of the contact contact and are as a section of the contact contact and the democratic lines and the democratic lines are for a first such as a section of the contact contact and the democratic lines are and the democratic lines are as a section of the contact and the democratic lines are as a section of the contact and the democratic lines are as a section of the contact and th

The control of the co

vee, dénieul studies have not been dese to demonstrate that we locking sortient lanses reduces the risk of developing catamets rays deserters. The Eye Gere Professional should be considited information.

The ADAM E GORDO Based Conduct Lens in relicated for the spicial correction of the ADAM E GORDO Based Contract of the contract

# ADVERSE REACTIONS The pasterit should be informed that the following problems may or

GENERAL FITTING GUIDELINES
A Patient Selection
Reports selected to sear these houses should be doosen based and The opening (Arm. 1800 and/or R.h.)

The opening (Arm. 1800 and/or R.h.)

There exists below controlled for other first report proby, southerd there exists the report proby, southerd the arm of the foreign of the arms the report proby, and the arms to arms the arms to arm to arm to arms the arms to arms the arms to arm the arms to arms the arms to arm to arm to arms the arms to arm the arms to arms the arms to arm to arm arms the arms the arms to arms the arms to arm to arms the arms the arms to arm to arms the arms the arms to arms the arms the arms to arms the arms the arms to arms the arms the arms to arms the arms the arms the arms the arms to arms the arms t

• Maling the Manager of the medical required by their mine one of the Maling of Manager I was a facility of the medical registration is prefer that the medical registration in the medical registration is prefer that the medical registration in the medical registration is prefer that the medical registration in the medical registration is prefer that the medical registration is prefer that the medical registration is prefer that the medical registration in the medical registration is prefer that the medical registration in the medical registration is prefer that the medical registration in the medical registration is prefer than the medical registration in the medical registration

V Vision of Unsuges,

- Loss of Walsen,

- C-C Ober Size Problems,

- C-C Ober Size Problems,

- G-C Ober Size Problems,

- G-C O

Ask to a stational information or thosis or the areator through or (fine or Asks to a stational information or thosis or stational information or enable to the stational enable to the stational enable to the stational enable to the stational or enable to the stational or enable to the stational enable to the stational or enable to the stational development and is enabled.

the design of the control of the con for A TERMATION Life. The Commission may provide these forms to write the A TERMATION Life. The Commission may provide these forms to a set the terman provide of commission may be compared to the terman to a set of the commission of commission may be considered to the Commission manufactured to the Commission of the context of the Commission of the Com

2. Others of a file limited lares of the foliation of the chaining the extensions: A file file by the stage of the lares of the report of the foliation of the chaining of the chaining of the file of the chaining of the ch

Q. Childo, M. & Shane Diffical and A family filling have used a high concernor of the following of membrane confliction increment and in a hist conjunctal hydroderic and mode after profession and design with the formal fill the since in Julyand interpolating in the Julyand and designment in the partners.

while their base curve in judged to be fitter or sheep fifting, the withern backet, builded be what face of bases of models to be a best for or desirated parts in temperature for the first and a broad in core from demonstrated depails, will fill not intern to a proposity content of position when the backet. It has a subsequent part of the first intern to a proposity content of position when the backet. It has a subsequently in the patient.

after innefing the new lens, the problem continues, the patient about the facultation and the CONTACT His CRINER APP CONTACT HIS OR HER APP ENDERSONAL.

The patient reports any problems, he or alse should be instructed to MMES, LY REMOYE, THE LERS. If the problem or discondust stops, the patient should docust the less and place a new healthers on the eye.

### **APPENDIX D:**

- Lens Fitting Characteristics
- Subject Reported Ocular Symptoms/Problems
- Front and Back Surface Lens Deposit Grading Procedure
- Determination of Distance Spherocylindrical Refractions
- Biomicroscopy Scale
- Keratometry Procedure
- Distance and Near Visual Acuity Evaluation
- Distance LogMAR Visual Acuity Measurement Procedure
- Patient Reported Outcomes
- White Light Lens Surface Wettability
- Visual Acuity Chart Luminance and Room Illumination Testing

# LENS FITTING CHARACTERISTICS

CR-6305, v4.0 Amendment 3.0














# SUBJECT REPORTED OCULAR SYMPTOMS/PROBLEMS

CR-6305, v4.0 Amendment 3.0














CR-6305, v4.0 Amendment 3.0 






# DETERMINATION OF DISTANCE SPHEROCYLINDRICAL REFRACTIONS



















# BIOMICROSCOPY SCALE

CR-6305, v4.0 Amendment 3.0













## KERATOMETRY PROCEDURE





# DISTANCE AND NEAR VISUAL ACUITY EVALUATION




















Page 2 of 3

CR-6305, v4.0 Amendment 3.0




## PATIENT REPORTED OUTCOMES





## WHITE LIGHT LENS SURFACE WETTABILITY







## VISUAL ACUITY CHART LUMINANCE AND ROOM ILLUMINATION TESTING














CR-6305, v4.0 Amendment 3.0




## PROTOCOL COMPLIANCE INVESTIGATOR(S) SIGNATURE PAGE

Protocol Number and Title: CR-6305: Design Validation of senofilcon A with New UV-blocking Additive

Version and Date: 4.0, Amendment 3.0 14 November 2018

I have read and understand the protocol specified above and agree on its content.

I agree to conduct this study according to ISO 14155, <sup>1</sup> GCP and ICH guidelines, <sup>2</sup> the Declaration of Helsinki, <sup>3</sup> United States (US) Code of Federal Regulations (CFR), <sup>4</sup> and the pertinent individual country laws/regulations and to comply with its obligations, subject to ethical and safety considerations. The Principal Investigator is responsible for ensuring that all clinical site personnel, including Sub-Investigators adhere to all ICH<sup>2</sup> regulations and GCP guidelines regarding clinical trials during and after study completion.

I will assure that no deviation from, or changes to the protocol will take place without prior agreement from the Sponsor and documented approval from the Institutional Review Board (IRB), except where necessary to eliminate an immediate hazard(s) to the trial participants.

I am responsible for ensuring that all clinical site personnel including Sub-Investigators adhere to all ICH<sup>2</sup> regulations and GCP guidelines regarding clinical trials during and after study completion.

All clinical site personnel involved in the conduct of this study have completed Human Subjects Protection Training.

I agree to ensure that all clinical site personnel involved in the conduct of this study are informed about their obligations in meeting the above commitments.

I shall not disclose the information contained in this protocol or any results obtained from this study without written authorization.

| Principal Investigator: | | |
|-------------------------|------------------------------------------|------|
| | Signature | Date |
| | | - |
| | Name and Professional Position (Printed) | |
| Institution/Site: | | |
| | Institution/Site Name | |
| | Institution/Site Address | |